| Division | : Worldwide Development |
|------------------|-------------------------------------|
| Information Type | : Reporting and Analysis Plan (RAP) |

| Title | porting and Analysis Plan for A aluate Safety, Tolerability, Pharmarmacodynamics of Single and R K3439171A, in a Randomized, Dolinded), Placebo- Controlled, Devaluate the Effect of Food on a K3439171A in Healthy Adult Pa | nacokinetics and Lepeat Oral Doses of Double-Blind (sponsor ose Escalation study and Single Oral Dose of |
|---|---|---|
| <b>Compound Number</b> | K3439171 | |
| <b>Effective Date</b> | Oct-2019 | |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 209275.
- This RAP is intended to describe the safety, tolerability, pharmacokinetic and pharmacodynamic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the reporting efforts, specifically Statistical Analysis Complete (SAC).

#### Author(s):

| Author | Date |
|---|---|
| Lead | 04-Oct- 2019 |
| Senior Statistician (FPD, Clinical Statistics) | |
| Co-Authors PPD | 04-Oct- 2019 |
| Clinical Pharmacologist (Clinical Pharmacology Modeling and Simulation) | 04-061-2019 |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited

# The GlaxoSmithKline group of companies

# **RAP Team Review Confirmations** (Method: E-mail)

| Reviewer | Date |
|---|---|
| Director, Clinical Statistics (FPD, Biostatistics) | 03-Oct- 2019 |
| Principal Statistician (FPD Clinical Statistics) | 04-Oct- 2019 |
| Director, Clinical Development (Disc Med) | 04-Oct- 2019 |
| Clinical Team Leader (FPD, Muscle Metabolism DPU) | 04-Oct- 2019 |
| Clinical Research Scientist (Global Clinical Sciences and Delivery, Clinical Projects and Quantitative Sciences) | 04-Oct- 2019 |
| Director, Clinical Development (Disc Med) | 04-Oct- 2019 |
| Medical Director, (Safety/ Pharmacovigilance) | 04-Oct- 2019 |
| Principal Data Manager (FPD, Global Clinical & Data Operations) | 04-Oct- 2019 |
| Biostatistics and Programming Manager (FPD, Biostatistics India) | 06-Oct- 2019 |

# Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma TMF eSignature)

| Approver | Date |
|---|---|
| Biostatistics and Programming Manager (FPD, Biostatistics India) | 09-Oct-2019 |
| Senior Manager - Biostatistics and Programming (FPD, Biostatistics India) | 09-Oct-2019 |

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTR | ODUCTIO | DN | 6 |
| 2. | SHM | MARY OF | KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | | es to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | | Objective(s) and Endpoint(s) | |
| | 2.3. | | Pesign | |
| | 2.4. | | al Hypotheses / Statistical Analyses | |
| 3. | PLAN | NED ANA | ALYSES | 12 |
| | 3.1. | | Analyses | |
| | 3.2. | | nalyses | |
| 4. | ANAL | YSIS PO | PULATIONS | 13 |
| | 4.1. | Protoco | l Deviations | 13 |
| 5. | | | IONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | | S | |
| | 5.1. | | reatment & Sub-group Display Descriptors | |
| | 5.2. | | e Definitions | 15 |
| | 5.3. | Other Conven | onsiderations for Data Analyses and Data Handling tions | 17 |
| ^ | OTUE | | | |
| 6. | | | LATION ANALYSES | |
| | 6.1. | Overvie | w of Planned Study Population Analyses | 18 |
| 7. | SAFE | | YSES | |
| | 7.1. | | e Events Analyses | |
| | 7.2. | | Laboratory Analyses | |
| | 7.3. | Other S | afety Analyses | 19 |
| 8. | PHAF | | NETIC ANALYSES | |
| | 8.1. | Primary | Pharmacokinetic Analyses | |
| | | 8.1.1. | | |
| | | | 8.1.1.1. Drug Concentration Measures | 20 |
| | | | 8.1.1.2. Derived Pharmacokinetic Parameters | <mark>20</mark> |
| | | 8.1.2. | Summary Measure | |
| | | 8.1.3. | Population of Interest | |
| | 8.2. | | ary Pharmacokinetic Analyses | |
| | | 8.2.1. | Endpoint / Variables | |
| | | | 8.2.1.1. Drug Concentration Measures | |
| | | | 8.2.1.2. Derived Pharmacokinetic Parameters | |
| | | 8.2.2. | Summary Measure | |
| | | 8.2.3. | Population of Interest | |
| | | 8.2.4. | Statistical Analyses / Methods | |
| | | | 8.2.4.1. Statistical Methodology Specification | 23 |

| | | 8.2.4.1.1. Statistical Methodology Specification for Part A (Single Dose) | 23 |
|---|---|---|---|
| | | 8.2.4.1.2. Statistical Methodology | |
| | | Specification for Part B | |
| | | Specification for Part C | |
| | 8.3. | Exploratory Pharmacokinetic Analyses | 28 |
| 9. | PHAR | MACOKINETIC (POPPK) ANALYSES | 29 |
| 10 | DHVD | MACODYNAMIC (AND / OR BIOMARKER) ANALYSES | 20 |
| 10. | 10.1. | | 29 |
| | 10.1. | 10.1.1. Endpoint / Variables | |
| | | 10.1.1.1. Drug Concentration Measures | |
| | | 10.1.2. Summary Measure | |
| | | 10.1.3. Population of Interest | |
| | | 10.1.4. Statistical Analyses / Methods | |
| | | 10.1.4.1. Statistical Methodology Specification | |
| | | 10.1.4.1.1. Statistical Methodology | |
| | | Specification for Part A (Single | |
| | | Dose) | 31 |
| | | 10.1.4.1.2. Statistical Methodology | |
| | | Specification for Part B (Repeat | |
| | | Dose) | 32 |
| 11 | DHVD | MACOKINETIC / PHARMACODYNAMIC ANALYSES | 33 |
| 11. | | ANIACONINE IIC / FIIANNIACOD INAINIIC ANAE I SES | |
| | REFE | RENCES | |
| 12. | | RENCES | 34 |
| 12. | APPE | RENCESNDICES | 34 |
| 12. | | NDICES | 34 |
| 12. | APPE<br>13.1. | RENCES NDICES Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population | 34<br>35 |
| 12. | APPE | NDICES Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population Appendix 2: Schedule of Activities | 34<br>35<br>35 |
| 12. | APPE<br>13.1.<br>13.2. | NDICES | 34<br>35<br>36<br>36 |
| 12. | APPE<br>13.1.<br>13.2.<br>13.3. | NDICES Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population Appendix 2: Schedule of Activities | 34<br>35<br>36<br>36 |
| 12. | APPE<br>13.1.<br>13.2. | NDICES | 35<br>35<br>36<br>36 |
| 12. | APPE<br>13.1.<br>13.2.<br>13.3. | NDICES | 34<br>35<br>36<br>36<br>73 |
| 12. | APPE<br>13.1.<br>13.2.<br>13.3. | NDICES Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population Appendix 2: Schedule of Activities 13.2.1. Protocol Defined Schedule of Events Appendix 3: Assessment Windows Appendix 4: Study Phases and Treatment Emergent Adverse Events 13.4.1. Study Phases | 34<br>35<br>36<br>36<br>73 |
| 12. | APPEI<br>13.1.<br>13.2.<br>13.3.<br>13.4. | NDICES | 34<br>35<br>36<br>36<br>73<br>74 |
| 12. | APPE<br>13.1.<br>13.2.<br>13.3. | NDICES Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population Appendix 2: Schedule of Activities 13.2.1. Protocol Defined Schedule of Events Appendix 3: Assessment Windows Appendix 4: Study Phases and Treatment Emergent Adverse Events 13.4.1. Study Phases for Concomitant Medication Appendix 5: Data Display Standards & Handling Conventions | 34353636737474 |
| 12. | APPEI<br>13.1.<br>13.2.<br>13.3.<br>13.4. | NDICES | 34<br>35<br>36<br>36<br>73<br>74<br>74<br>75 |
| 12. | APPEI<br>13.1.<br>13.2.<br>13.3.<br>13.4. | NDICES Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population Appendix 2: Schedule of Activities 13.2.1. Protocol Defined Schedule of Events Appendix 3: Assessment Windows Appendix 4: Study Phases and Treatment Emergent Adverse Events 13.4.1. Study Phases 13.4.1. Study Phases for Concomitant Medication Appendix 5: Data Display Standards & Handling Conventions 13.5.1. Reporting Process 13.5.2. Reporting Standards | 34<br>35<br>36<br>36<br>73<br>74<br>74<br>75<br>75 |
| 12. | APPEI<br>13.1.<br>13.2.<br>13.3.<br>13.4. | NDICES Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population. Appendix 2: Schedule of Activities 13.2.1. Protocol Defined Schedule of Events. Appendix 3: Assessment Windows Appendix 4: Study Phases and Treatment Emergent Adverse Events 13.4.1. Study Phases 13.4.1.1. Study Phases for Concomitant Medication. Appendix 5: Data Display Standards & Handling Conventions. 13.5.1. Reporting Process 13.5.2. Reporting Standards. 13.5.3. Reporting Standards for Pharmacokinetic. | 343536367374747575 |
| 12. | APPEI<br>13.1.<br>13.2.<br>13.3.<br>13.4. | NDICES Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population Appendix 2: Schedule of Activities 13.2.1. Protocol Defined Schedule of Events Appendix 3: Assessment Windows Appendix 4: Study Phases and Treatment Emergent Adverse Events 13.4.1. Study Phases 13.4.1. Study Phases for Concomitant Medication Appendix 5: Data Display Standards & Handling Conventions 13.5.1. Reporting Process 13.5.2. Reporting Standards | 34353636737474757575 |
| 12. | APPEI<br>13.1.<br>13.2.<br>13.3.<br>13.4. | NDICES Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population | 3435363673747475757576 |
| 12. | APPEI<br>13.1.<br>13.2.<br>13.3.<br>13.4. | NDICES Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population | 3435363673747475757579 |
| 12. | APPEI<br>13.1.<br>13.2.<br>13.3.<br>13.4. | NDICES Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population Appendix 2: Schedule of Activities 13.2.1. Protocol Defined Schedule of Events Appendix 3: Assessment Windows Appendix 4: Study Phases and Treatment Emergent Adverse Events 13.4.1. Study Phases 13.4.1.1. Study Phases for Concomitant Medication Appendix 5: Data Display Standards & Handling Conventions 13.5.1. Reporting Process 13.5.2. Reporting Standards 13.5.3. Reporting Standards for Pharmacokinetic Appendix 6: Derived and Transformed Data 13.6.1. General 13.6.2. Study Population | 343536367374747575757979 |
| 12. | APPEI<br>13.1.<br>13.2.<br>13.3.<br>13.4. | NDICES Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population. Appendix 2: Schedule of Activities 13.2.1. Protocol Defined Schedule of Events. Appendix 3: Assessment Windows. Appendix 4: Study Phases and Treatment Emergent Adverse Events. 13.4.1. Study Phases for Concomitant Medication. Appendix 5: Data Display Standards & Handling Conventions. 13.5.1. Reporting Process. 13.5.2. Reporting Standards. 13.5.3. Reporting Standards for Pharmacokinetic. Appendix 6: Derived and Transformed Data 13.6.1. General. 13.6.2. Study Population. 13.6.3. Safety | 3435363673747475757576798081 |

#### CONFIDENTIAL

| | 13.7.2. | Handling of Missing Data | .83 |
|---|---|---|---|
| | | 13.7.2.1. Handling of Missing and Partial Dates | |
| | | 13.7.2.2. Handling of PK Concentration Data | |
| | | 13.7.2.3. Handling of Missing Data for Statistical | |
| | | Analysis | .84 |
| 13.8. | Appendix | x 8: Values of Potential Clinical Importance | .85 |
| | | Laboratory Values | |
| | 13.8.2. | ECG | .86 |
| | 13.8.3. | Vital Signs | .86 |
| 13.9. | Appendix | x 9: Population Pharmacokinetic (PopPK) Analyses | .87 |
| 13.10. | Appendix | x 10: Pharmacokinetic / Pharmacodynamic Analyses | .88 |
| 13.11. | Appendix | x 11: Abbreviations & Trade Marks | .89 |
| | 13.11.1. | Abbreviations | .89 |
| | 13.11.2. | Trademarks | .90 |
| 13.12. | Appendix | x 12: List of Data Displays | .91 |
| | | Data Display Numbering | |
| | 13.12.2. | Mock Example Shell Referencing | .91 |
| | 13.12.3. | Deliverables | .92 |
| | 13.12.5. | Safety Tables | . 96 |
| | | Safety Figures | |
| | 13.12.7. | Pharmacokinetic Tables | 113 |
| | 13.12.8. | Pharmacokinetic Figures | 116 |
| | 13.12.9. | Pharmacodynamic (and / or Biomarker) Tables | 118 |
| | 13.12.10 | .Pharmacodynamic (and / or Biomarker) Figures | 123 |
| | | .ICH Listings | |
| | 13.12.12 | .Non-ICH Listings | 155 |
| | | Other Listings | |
| 13.13. | Example | Mock Shells for Data Displays | 158 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 209275:

| Revision Chronology: | | |
|---|---|---|
| 2018N361438_00 | 03-JUL-2018 | Original |
| 2018N361438_01 | 27-AUG-2018 | Updates to the PK exposure limits for Parts A and B, stopping criteria, and safety review language have been modified based on FDA recommendations. Day -2 has also been removed from Part C of the SoA as it is not necessary. Information around Holter Monitoring has been altered to reflect the intent of collecting but not analyzing Holter Monitoring data in this study. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

- **Detail to Include**: Outline & fully justify (where applicable) changes to the planned protocol analysis.
  - o If there are no changes or deviations from the protocol, then specify within this section.

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Analysis population: Enrolled population has been removed from the population definitions. | Analysis population: Screened population definition has been added to the population definitions. | More specific definition<br>according to the new RAP<br>template |
| Analysis population: Evaluable population has been removed from the population definitions. | • | This population will be equivalent to the PK/PD population which are already included |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To assess the safety and tolerability of GSK3439171A following single and repeat doses in healthy participants | Adverse events (AE), Serious Adverse Events (SAE), clinical laboratory values, vital signs, and electrocardiograms (ECG) |
| To characterize the PK of GSK3439171A, following single and repeat doses in healthy participants | Derived PK parameters for GSK3439171A including area under the plasma drug concentration versus time curve (AUC(0-t), AUC(0-inf), maximum observed plasma drug concentration (Cmax), time to maximum observed plasma drug concentration (tmax), and apparent terminal half-life (t1/2) as appropriate |
| Secondary Objectives | Secondary Endpoints |
| To assess the effect of food on the PK of GSK3439171A following an oral dose in healthy participants | Derived PK parameters for GSK3439171A including area under the plasma drug concentration versus time curve (AUC(0-t), AUC(0-inf), maximum observed plasma drug concentration (Cmax), time to maximum observed plasma drug concentration (tmax), and apparent terminal half-life (t1/2) as appropriate |
| To assess preliminary dose proportionality of GSK3439171A following single and repeat oral doses, as data permit | AUC(0-t), AUC(0-inf), and Cmax following single dose and AUC(0-τ) and Cmax following repeat dose for the assessment of dose proportionality |
| To examine the extent of accumulation and achievement of steady-state following repeat oral doses of GSK3439171A, as data permits | <ul> <li>Determine observed accumulation based on AUC(Ro) and Cmax (RCmax) and determine the steadystate ratio (Rss)</li> <li>Trough plasma concentrations at the end of the dosing interval (Cτ) collected pre-dose for repeat doses 12, 13 and 14* to assess the achievement of steady-state of GSK3439171A</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate the PD properties of GSK3439171A | Levels of mediators on prostaglandin and/or inflammatory metabolic pathways such as, but not limited to, PGD2, and PGE2. |
| To assess the effect of GSK3439171A on QTc in healthy adult volunteers | Holter monitor data collection and storage for evaluation of the correlation between plasma levels of GSK3439171A and changes in the QTc interval in the future, if appropriate |
| To evaluate additional biomarkers of GSK3439171A target | Levels of change in novel biomarkers in blood, muscle, or urine, such as, but not limited to, urine |

| Objectives | Endpoints |
|---|---|
| engagement after single and repeat | tetranor PGDM and PGEM (tPGDM, tPGEM), |
| doses. | PGD2, and PGE2 |
| To investigate the plasma, urinary | GSK3439171-related material in plasma, urine and |
| and biliary (Part B) metabolic | bile |
| pathways of GSK3439171A in | |
| healthy subjects | |
| * 12, 13 and 14 changed to 6,7,9,10, 11, 15,16, and 17 | |

# 2.3. Study Design

#### Overview of Study Design and Key Features Part A: Single Ascending Dose Treatment Period Screening (~30 days prefirst dose) Cohort A1, n=9 (6A:3P, Cohort A2, n=9 (6A:3P, Cohort A3, n=9 (6A:3P. 3 participants / sequence PBO PBO PBO Dose 9 Dose 2 Dose 3 Dose 5 Dose 6 Dose 8 Dose 1 PBO Dose 3 **PBO** Dose 6 Dose 1 PBO P80 Dose 2 Dose 4 Dose 5

Within a cohort, participants will be randomized to one of 3 treatment sequences such that each participant receives 2 active doses and 1 placebo dose resulting in each active dose being administered to 6 participants and placebo to 3 participants

- Starting dose (Dose 1) = 5 mg
- Subsequent dose escalations will be determined based on safety and PK data
- Maximum predicted dose = 500 mg (Genotoxic Risk Assessment Limit= 3000mg)
- Washout= 7 days or 5 half-lives, whichever is longer
- = Dose escalation meeting

PBO= Placebo

\*Note: dosing strategy is for illustrative purposes and does not represent the randomization strategy

### Part B: Single and Repeat Dose 14-day dose-rising



Doses will be selected based on safety, tolerability and PK data from Part A

= Dose escalation meeting

#### Part C: Food Effect



- 7-day or 5 half-lives (whichever is longer) washout period/ participant crossover to fasted/fed arm

| Overview of St | udy Design and Key Features |
|---|---|
| Design<br>Features | Part A is a randomized, double blind, placebo-controlled, crossover, single dose escalation study in healthy participants. Participants will be randomized to placebo or active study intervention groups after screening. |
| | Part B is a randomized, double blind, placebo-controlled, parallel group, repeat dose escalation study in healthy participants. Participants will be randomized to placebo or active study intervention groups after screening. |
| | <ul> <li><u>Part C</u> is a randomized, open label, crossover, food effect study in<br/>healthy participants. Participants will be randomized to fed or fasted<br/>groups after screening.</li> </ul> |
| Dosing | <ul> <li>Part A: Each participant will participate in 3 dosing periods and will receive 2 doses of GSK3439171A and 1 dose of placebo in a randomized fashion. There will be an approximately 7 day (or 5 half-lives, whichever is longer) washout period between dosing in each session. Each active dose level will be administered initially to a smaller group of participants (1on active and 1 on placebo) and will be followed clinically for 48 hr (or 5 half-lives, whichever is longer) to allow for adequate observation of safety. If no acute safety issues are observed in this smaller group of sentinel participants, then the remaining participants (approximately 5 participants on active and 2 participants on placebo) will receive the dose.</li> <li>Part B: In each cohort of Part B of the study, approximately twelve participants will be randomized to either one dose level of GSK3439171A or placebo according to a randomization schedule prepared prior to the start of the study. The study will be conducted sequentially starting with Dose 1 Cohort B1. Participants will receive a single dose followed by a 48 hr assessment period and then will receive daily repeat doses until the end of the study.</li> <li>Part C: In this crossover design, approximately 12 participants will take part in two periods with dosing in each period separated by approximately 7 days (or 5 half-lives of the study intervention, whichever is longer). In each study session, participants will be admitted to the clinical unit and receive a single dose of GSK3439171A either in the fasted state or after a high fat meal.</li> </ul> |
| Time & Events | Refer to Appendix 2: Schedule of Activities |
| Treatment<br>Assignment | Participants will be randomized to receive study intervention. Randomization schedule generated using RandAll NG prior to the study by the Clinical Statistics Department at GSK will be sent to the site and the site pharmacist randomizes the participants according to the randomization schedule. Investigators and all site staff with the exception of the pharmacy staff will remain blinded to each participant's assigned study intervention throughout the course of the study. • Part A: approximately 9 participants in each cohort will be randomized to one of 3 treatment sequences for 3 cohorts. Within each period, allocation of active (A) to placebo (P) treatment will be 2:1. Within a cohort, an increasing dose of GSK3439171A will be administered in each period. • Part B: In each cohort of, approximately 12 participants will be randomized to receive either GSK3439171A or placebo in a parallel design using a 3:1 allocation ratio. |
| | Part C: Approximately 12 participants will be randomized 1:1 to receive |

| Overview of St | Overview of Study Design and Key Features |
|---|---|
| | GSK3439171A in one of two treatment sequences (Fed then Fasted or Fasted then Fed). |
| Interim<br>Analysis | There will be no formal statistical interim analysis. However, preliminary safety, PK, and PD/biomarker data will be reviewed in-stream by the GSK study team members prior to each dose escalation. Data for these reviews will be cumulative and can include individual participant data, summaries by treatment group and graphical displays. This is a sponsor unblinded trial and GSK staff will be unblinded for these reviews. |

# 2.4. Statistical Hypotheses / Statistical Analyses

The primary objectives of this study are to evaluate safety and tolerability of single and repeat doses of GSK3439171A and to characterize the PK of GSK3439171A. No formal statistical hypotheses will be tested. Descriptive statistics will be used to assess safety and tolerability objectives. Treatment comparisons with placebo will be based on review of descriptive statistics and individual participant data. An estimation approach will be used to address the PK objectives where point estimates and corresponding 90% confidence intervals (CIs) will be constructed as appropriate for the assessment of dose proportionality, steady-state, time invariance and food effect.

#### 3. PLANNED ANALYSES

# 3.1. Interim Analyses

There will be no formal statistical interim analysis. However, preliminary safety, PK, and PD/biomarker data will be reviewed in-stream by the GSK study team members and investigational site (PAREXEL) team prior to each dose escalation. This data review is conducted in two steps: First GSK staff will review the unblinded data, as this is a sponsor unblinded trial and then the blinded data will be presented to investigational site team in another meeting. Data for these reviews will be cumulative and can include individual participant data, summaries by treatment group and graphical displays.

Preliminary results from available safety data may be reported prior to database freeze for the purposes of safety review by GSK, and where required by regulatory bodies. Other selected preliminary data may be unblinded and reported prior to database freeze for internal decision making. In each case described above, the study will not be officially unblinded and access to the randomization will be restricted.

After completing Part A and cohort 1&2 for Part B there was a safety review of the unblinded data to decide if higher dose can be administered for cohort 3 in Part B. Summaries and figures for Clinical chemistry, Hematology and Hormone level were created for the safety review (The displays that were created are indicated in list of data displays). Unblinded results were produced for an IB update, which was a subset of Study population, Safety and PK concentration displays, more details of the results submitted will be documented in IB update documentation.

Summaries and graphical displays for in-stream reviews will not be provided by Statistics and Programming and as such, no details on these summaries are provided in the RAP.

# 3.2. Final Analyses

Final analyses will be reported when all subjects in all cohorts have completed their final scheduled visits and the following sequential steps have occurred:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | Screen Failures |
| Randomized | All participants who were randomized | Study Population |
| Safety | All participants who take at least 1 dose of study intervention. Participants will be analyzed according to the intervention they actually received. | Study Population<br>Safety |
| PK | Participants in the Safety population for whom a PK sample was taken and analyzed for GSK3439171A and result reported | PK |
| PD | Participants in the Safety population with at least one PD measure. | PD/Biomarker |

Refer to Appendix 12: List of Data Displays which details the population used for each display. Metabolite ID work will be reported in a separate GSK report

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the ClinBase.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

- There are no planned adjustments made for multiple centres in this study.
- There are no planned adjustments for multiple comparisons or multiplicity.

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG | Data Displays fo | or Reporting |
| Code | Description | Description | Order in TLF |
| Part A | | | |
| D1 | GSK3439171A Dose 1 | 5 mg | 2 |
| D2 | GSK3439171A Dose 2 | 10 mg | 3 |
| D3 | GSK3439171A Dose 3 | 30 mg | 4 |
| D4 | GSK3439171A Dose 4 | 60 mg | 5 |
| D5 | GSK3439171A Dose 5 | 120 mg | 6 |
| D6 | GSK3439171A Dose 6 | 180 mg | 7 |
| PA | Placebo Part A | Placebo | 1 |
| Part B | | | |
| DD1 | GSK3439171A R1 mg QD or<br>BID | 5 mg | 10 |
| DD2 | GSK3439171A R2 mg QD or<br>BID | 11 mg | 11 |
| DD3 | GSK3439171A R3 mg QD or<br>BID | 40 mg | 12 |
| PB | Placebo Part B | Placebo | 8 |
| PB3 | Placebo Part B Cohort 3 | Placebo Cohort 3 | 9 |

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code | Description | Description Order in TLF | |
| Part C | Part C | | |
| C1 | GSK3439171A fasted | 60 mg Fasted | 13 |
| C2 | GSK3439171A fed | 60 mg Fed | 14 |

Note: If additional dose levels are explored in either Part A or B, then they will follow in a sequential order in the table

Treatment comparisons will be displayed as follows using the descriptors as specified:

- 1. Day 17 vs Day 1 (e.g.; Ro, RCmax and Rss)
- 2. Dose X.X mg vs Placebo
- 3. Repeat Dose X.X mg vs Placebo
- 4. Fasted vs Fed

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. For the parameters having multiple assessments, mean value of the assessments will be considered as baseline value.

#### **Baseline Definitions – Part A**

| Parameter | Study Assessments Considered as Baseline | | | | Baseline Used |
|---|---|---|---|---|---|
| | Screening | Day -2 | Day -1 | Day 1 (Pre-<br>Dose) | in Data Display |
| <b>Safety Assessments</b> | | | | | |
| Lab results, 12-<br>lead<br>Electrocardiogram<br>(ECG) & Vital<br>Signs | X | X | | X | Day 1 |
| Routine Urinalysis | X | | | X | Day 1 |
| Telemetry | | | | X | Day 1<br>30 min (±10<br>min) |
| Pharmacodynamics parameters | | | X | X | Day -1 # |

# Postdose value will be collected on intervals 0-2, 2-4, 4-6, 6-8, 8-12 and 12-24 hr. Time matched predose value for each of these intervals (24-22, 22-20, 20-18, 18-16, 16-12 and 12-0 respectively), predose aggregate value of 24-12hr (for post dose aggregate of 0-12 hrs) and predose aggregate value of 12-0 hr (for post dose aggregate of 12-24 hrs) will be considered as baseline for different pharmacodynamic parameters

#### **Baseline Definitions - Part B**

| Parameter | Study A | Assessments | Baseline Used in | | |
|---|---|---|---|---|---|
| | Screening | Day -2 | Day -1 | Day 1 (Pre-<br>Dose) | Data Display |
| Safety Assessments | | | | | |
| Lab results | X | X | X | X | Day 1 |
| Hormone<br>monitoring | | | X | | Day -1† |
| Routine Urinalysis,<br>12-lead<br>Electrocardiogram<br>(ECG) & Vital<br>Signs | Х | X | | X | Day 1 |
| Telemetry | | | | X | Day 1<br>30 min (±10<br>min) |
| Pharmacodynamics parameters | | | X | X | Day -1 # |
| Blood sampling for<br>metabolite<br>profiling | | | | X | Day 1 (pre-<br>dose) |
| Muscle Biopsy | | | X | | Day -1 |

<sup>&</sup>lt;sup>†</sup> There will be 2 individual baseline values (samples from midnight and 9am) for ACTH and Cortisol hormones. Both values may be used to calculate change from baseline for post dose measurements.

<sup>#</sup> Postdose value will be collected on intervals 0-2, 2-4, 4-6, 6-8, 8-12 and 12-24hr. Time matched predose value for each of these intervals (24-22, 22-20, 20-18, 18-16, 16-12 and 12-0 respectively), predose aggregate value of 24-12hr (for post dose aggregate of 0-12 hrs) and predose aggregate value of 12-0 hr (for post dose aggregate of 12-24 hrs) will be considered as baseline for different pharmacodynamic parameters

#### **Baseline Definitions – Part C**

| Parameter | Study Asse | Study Assessments Considered as Baseline | | |
|---|---|---|---|---|
| | Screening | Screening Day -1 Day 1 (Pre-Dose) | | in Data Display |
| Safety Assessments | | | | |
| Lab results, 12-lead<br>Electrocardiogram<br>(ECG) & Vital Signs | X | | X | Day 1 |
| Routine Urinalysis | X | | X | Day 1 |
| Telemetry | | | X | Day 1<br>30 min (±10<br>min) |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 13.3 | Appendix 3: Assessment Windows |
| 13.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 13.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 13.6 | Appendix 6: Derived and Transformed Data |
| 13.7 | Appendix 7: Reporting Standards for Missing Data |
| 13.8 | Appendix 8: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the randomised population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 12: List of Data Displays.

# 7. SAFETY ANALYSES

The safety analyses will be based on the safety population, unless otherwise specified.

Descriptive statistics will be used to assess safety and tolerability objectives. No formal statistical analyses of safety data are planned. Data will be summarized according to GSK Integrated Data Standards Library (IDSL) standards for Part A, Part B and Part C separately. In addition, individual participant data will be reviewed. Treatment comparisons with placebo will be based on review of descriptive statistics and individual participant data.

# 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious adverse events (SAEs) and other significant AEs will be based on GSK Core Data Standards.

## 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, Liver chemistries and Hormone assessment tests will be based on GSK Core Data Standards. Hormone assessment tests will be done in Part B only and all the other laboratory evaluations will be done for all the 3 parts (A, B & C) of the study.

# 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs vital signs and Telemetry will be based on GSK Core Data Standards, unless otherwise specified.

#### 8. PHARMACOKINETIC ANALYSES

# 8.1. Primary Pharmacokinetic Analyses

## 8.1.1. Endpoint / Variables

Pharmacokinetic parameters will be determined from the plasma concentration-time data, as data permits.

PK parameters: Maximum observed blood concentration (Cmax), time to Cmax (tmax), area under the plasma concentration-time curve [AUC(0-t), AUC(0-24), AUC(0-inf) and AUC(0- $\tau$ )], Pre-dose observed concentration (C $\tau$ ), apparent terminal phase half-life (t1/2) will be determined, as data permit.

#### 8.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 13.5.3. Reporting Standards for Pharmacokinetic)

#### 8.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix 64. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

 Table 2
 Derived Pharmacokinetic Parameters (Primary end points)

| Parameter | Parameter Description | Part A | Part B | Part C |
|---|---|---|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) which will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. | X | X <sup>1</sup> | X |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity calculated as $AUC(0-\infty)=AUC(0-t)+C(t)/lambda_z$ | X | X <sup>1</sup> | X |
| AUC(0-24) | Area under the concentration-time curve from time zero to 24 hours post-dose which will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. | X | X <sup>1,2</sup> | |

| Parameter | Parameter Description | Part A | Part B | Part C |
|---|---|---|---|---|
| tmax | Time to reach Cmax, determined directly | X | $X^{1,2}$ | X |
| | from the concentration-time data. | | | |
| t1/2 | Apparent terminal half-life will be | X | $X^{1,2}$ | X |
| | calculated as: | | | |
| | $t^{1/2} = \ln 2 / \text{lambda}_z$ | | | |
| Ae | Urinary excretion of unchanged drug | | $X^{1,2}$ | |
| Clr | Renal clearance | | $X^{1,2}$ | |
| Fe | Fraction of the dose excreted in the urine | | $X^{1,2}$ | |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. | X | X <sup>1,2</sup> | X |
| Ст | Pre-dose observed concentration (trough) for repeat doses on Days 6,7,9,10, 11, 15,16, and 17 (6, 7, 9 & 10 for 7 day repeat dosing) which will be obtained directly from the concentration-time data. | | X <sup>1,2</sup> | |

Additional parameters may be calculated as required.

Lambda\_z is the terminal phase rate constant.

# 8.1.2. Summary Measure

Pharmacokinetic data will be presented in graphical and/or tabular form and will be summarized descriptively by dose group for each study part separately.

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 13.5.3. Reporting Standards for Pharmacokinetic)

Pharmacokinetic analysis will be the responsibility of the Clinical Pharmacology Modelling and Simulation Department, CPMS, GlaxoSmithKline and Statistical analyses of the pharmacokinetic parameter data will be the responsibility of Clinical Statistics & Programming, GlaxoSmithKline.

## 8.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

# 8.2. Secondary Pharmacokinetic Analyses

### 8.2.1. Endpoint / Variables

Observed accumulation ratio AUC(Ro), predicted accumulation ratio AUC(Rp), observed accumulation ratio for Cmax (RCmax) and steady state ratio (Rss).

<sup>&</sup>lt;sup>1</sup>Determined for dose 1

<sup>&</sup>lt;sup>2</sup>Determined at SS (following 14 days of consecutive dosing)

#### 8.2.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 13.5.3 Reporting Standards for Pharmacokinetic)

#### 8.2.1.2. Derived Pharmacokinetic Parameters

 Table 3
 Derived Pharmacokinetic Parameters (Secondary end points)

| Parameter | Parameter Description | Part A | Part B | Part C |
|---|---|---|---|---|
| % AUCex | The percentage of AUC $(0-\infty)$ obtained by extrapolation (%AUCex) will be calculated as: AUC $(0-\infty)$ - AUC $(0-t)$ /AUC $(0-\infty)$ x 100 | X | X | X |
| AUC(Ro) | Observed accumulation ratio (Ro) for AUC will be calculated as follows: Day 17 AUC(0- $\tau$ )/Day 1 AUC(0- $\tau$ ) | | X <sup>1</sup> | |
| AUC(Rp) | Predicted accumulation ratio will be calculated as follows: Day 1 AUC(0- ∞)/Day 1 AUC(0- 24) | Х | X <sup>1</sup> | Х |
| Rss | Steady state accumulation ratio (Rss) will be calculated as follows: Day 17 AUC(0- τ)/Day 1 AUC(0-∞) | | X <sup>1</sup> | |
| RCmax | Observed accumulation ratio for Cmax (Rcmax) will be calculated as follows: Day 17 Cmax/Day 1 Cmax | | X <sup>1</sup> | |

<sup>&</sup>lt;sup>1</sup>Day 10 AUC will be considered instead of Day 17 for the reduced treatment period cohort (Part B cohort3).

#### 8.2.2. Summary Measure

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 13.5.2. Reporting Standards for Pharmacokinetic)

#### 8.2.3. Population of Interest

The secondary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

#### 8.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.2.1.2 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 8.2.4.1. Statistical Methodology Specification

### 8.2.4.1.1. Statistical Methodology Specification for Part A (Single Dose)

### Pharmacokinetic Statistical Analyses – ANOVA – Single Dose (Part A)

#### **Endpoint / Variables**

AUC(0-t), AUC(0-24), AUC(0- $\infty$ ), Cmax, C $\tau$ , t1/2, AUC(Rp)

### **Model Specification**

Actual value of t1/2 and loge-transformed values of rest of the endpoints will be statistically analyzed using Mixed Model (MM) ANOVA.

- Fixed effect: dose
- Random effect: Subject

An unstructured covariance structure for the G matrix will be used.

- If this model fails to converge, alternative covariance structures may be considered.
- Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.

Analyses will be done with the MIXED Procedure in SAS, using the Kenward-Roger option to estimate denominator degrees of freedom and standard errors

#### **Model Checking & Diagnostics**

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold.

#### **Model Results Presentation**

LSmeans and 90% CI are estimated for each dose as well as overall estimate of within-subject CV

Note: AUC(0-t) is only reported when AUC(0-∞) is not reportable

# Pharmacokinetic Statistical Analyses - Dose Proportionality (Power Model) - Single Dose (Part A)

#### **Endpoint / Variables**

Single Dose: AUC(0-t), AUC(0-∞) and Cmax

#### **Model Specification**

Will be statistically analyzed using the power model

 $y = \alpha^* dose\beta$ 

Where y =PK parameter being analyzed and  $\alpha$ = subject

Loge transformed data will be analyzed by fitting the following terms in the mixed effect model:

- Fixed effect: loge (dose)
- Random effect: Subject (Intercept only)

### **Model Checking & Diagnostics**

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold.

#### **Model Results Presentation**

Estimates of the mean slopes of log<sub>e</sub> (dose) will be reported along with corresponding 90% confidence intervals (slope≈1 implies dose proportionality)

Note: AUC(0-t) is only reported when AUC(0- $\infty$ ) is not reportable

#### 8.2.4.1.2. Statistical Methodology Specification for Part B

# Pharmacokinetic Statistical Analyses – ANOVA (Accumulation & Time Invariance) – Repeat Dose (Part B)

#### **Endpoint / Variables**

AUC(0- $\tau$ ), AUC(0- $\infty$ ), Cmax, C $\tau$ , AUC Rss, t1/2, AUC (Ro), RCmax

#### Model Specification

Actual value of t1/2 and loge-transformed values of all other will be statistically analyzed using Mixed Model (MM) ANOVA.

- Fixed effect: day, dose, day\*dose
- Random effect: Subject

An unstructured covariance structure for the G matrix will be used.

- If this model fails to converge, alternative covariance structures may be considered.
- Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.

Analyses will be done with the MIXED Procedure in SAS, using the Kenward-Roger option to estimate denominator degrees of freedom and standard errors

#### **Model Checking & Diagnostics**

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold.

#### **Model Results Presentation**

LSmeans and 90% CI are estimated for each dose as well as overall estimate of within-subject CV. For AUC(0- $\tau$ ), Cmax and AUC-Rss, estimates of ratio of Day 17to Day 1 will be evaluated for each dose by exponentiating the difference in least squares means (Day 17– Day 1) and the associated 90% CI. Such that ratios of Day 17 to Day 1 for AUC(0- $\tau$ ), Cmax and AUC-Rss provide estimates of Ro, RCmax and Rss, respectively

Note: For AUC-Rss, Day 17 AUC(0- $\tau$ ) and Day 1 AUC(0- $\infty$ ) should be considered.

Note: Day 10 values will be considered instead of Day 17 for the reduced treatment period cohort (cohort 3)

# Pharmacokinetic Statistical Analyses - Dose Proportionality (Power Model) - Repeat Dose (Part B)

#### **Endpoint / Variables**

Repeat Dose: AUC(0- $\tau$ ) and Cmax

### **Model Specification**

Will be statistically analyzed using the power model

 $y = \alpha^* dose\beta$ 

Where y =PK parameter being analyzed and  $\alpha$ = subject

Loge transformed data will be analyzed by fitting the following terms in the mixed effect model:

- Fixed effect: log<sub>e</sub> (dose)
- Random effect: Subject (Intercept only)

#### **Model Checking & Diagnostics**

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.

Non-parametric analyses will be conducted if the normality assumption does not hold.

#### **Model Results Presentation**

Estimates of the mean slopes of log<sub>e</sub> (dose) will be reported along with corresponding 90% confidence intervals (slope≈1 implies dose proportionality)

#### Pharmacokinetic Statistical Analyses - Achievement of Steady State - Repeat Dose (Part B)

#### **Endpoint / Variables**

Trough plasma concentrations at the end of the dosing interval ( $C\tau$ ) for repeat doses Days 6,7,9,10, 11, 15,16, and 17 (6, 7, 9 & 10 for reduced treatment period cohort)

#### **Model Specification**

Log<sub>e</sub>-transformed values of the endpoint will be statistically analyzed separately by dose using Mixed Model (MM) ANOVA.

- Fixed effect: day as continuous variable, dose, day\*dose
- Random effect: Subject

An unstructured covariance structure for the G matrix will be used.

- In the event that this model fails to converge, alternative covariance structures may be considered.
- Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.

Analyses will be done with the MIXED Procedure in SAS, using the Kenward-Roger option to estimate denominator degrees of freedom and standard errors

#### **Model Checking & Diagnostics**

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold.

#### **Model Results Presentation**

The coefficient for the slope of the day effect on the log-scale will be used to evaluate steady state for each dose. The 90% confidence intervals for the slope will be calculated.

Steady-state will be assessed visually by plotting trough concentration levels, CT, collected premorning dose versus collection day by dose.

#### 8.2.4.1.3. Statistical Methodology Specification for Part C

#### Pharmacokinetic Statistical Analyses - Food Effect -Single Dose (Part C)

#### **Endpoint / Variables**

AUC(0-t), AUC(0- $\infty$ ), Cmax and t1/2

#### **Model Specification**

 $Log_e$ -transformed values of AUC(0-t) and AUC(0- $\infty$ ) and actual value of t1/2 will be statistically analyzed using Mixed Model (MM) ANOVA.

- Fixed effect: period, treatment(fed/fasted)
- Random effect: Subject

An unstructured covariance structure for the G matrix will be used.

- If this model fails to converge, alternative covariance structures may be considered.
- Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.

Analyses will be done with the MIXED Procedure in SAS, using the Kenward-Roger option to estimate denominator degrees of freedom and standard errors

#### **Model Checking & Diagnostics**

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold.

#### **Model Results Presentation**

Point estimates for the differences in means (GSK3439171A fed – GSK3439171A fasted) and corresponding 90% CIs will be constructed from the least squares means, using the residual variance. These will then be back-transformed to provide point estimates and corresponding 90% CIs for the ratio of geometric means fed:fasted.

#### Endpoint(s)

Tmax

Note: This endpoint will not be log transformed for analysis

#### Model Specification

Wilcoxon matched pair test

#### Model Results Presentation

Point estimate and 90% confidence interval for the median difference (fed – fasted)

Note: AUC(0-t) is only reported when AUC(0- $\infty$ ) is not reportable Population

# 8.3. Exploratory Pharmacokinetic Analyses

If data permits, PK data of metabolites will be analyzed in the similar way as for drug substance and similar output will be generated.

# 9. PHARMACOKINETIC (POPPK) ANALYSES

PopPK will be performed under a separate RAP and will be reported separately.

# 10. PHARMACODYNAMIC (AND / OR BIOMARKER) ANALYSES

# 10.1. Exploratory Pharmacodynamic and Biomarker Analyses

# 10.1.1. Endpoint / Variables

Following table describes the pharmacodynamic/biomarker end points:

| Parameter | meter Parameter Description/Derivation | | |
|---|---|---|---|
| PGD2 | | | X |
| PGE2 | | | Χ |
| Creatinine # | | Х | Χ |
| tPGDM# | | Х | Χ |
| tPGEM# | | Х | Χ |
| 6-keto-PGF1A | | | Χ |
| PGF2A | | | Χ |
| TXB2 | | | Χ |
| Creatinine corrected data for tPGDM and tPGEM # | Three versions of data to be considered: 1.Raw data(mass) 2. Aggregated data 0-12hrs 3. Aggregated data 12-24hr 4. Aggregated data 24-48hrs Each version of data(mass) divided by time matched creatinine(mass) | Х | X |
| Baseline corrected<br>urinary tetranor data<br>for tPGDM and<br>tPGEM # | Post dose data divided by time matched baseline data Three versions of data to be considered: 1.Creatinine corrected raw data 2. Creatinine corrected aggregated data 0-12hrs 3. Creatinine corrected aggregated data 12-24hrs | X | X |
| Baseline corrected urinary tetranor data for creatinine # | ary tetranor data data | | |

| Parameter | Parameter Description/Derivation | Part A | Part B |
|---|---|---|---|
| Placebo corrected<br>data for tPGDM and<br>tPGEM# | Creatinine corrected data from active dose divided by time matched placebo data and then find ratio to baseline. Three versions of data to be considered: 1.Creatinine corrected raw data 2. Creatinine corrected aggregated data 0-12hrs 3. Creatinine corrected aggregated data 12-24hrs | X | |
| Placebo corrected data for creatinine # | Data from active dose divided by time matched placebo data and then find ratio to baseline. Three versions of data to be considered: 1.Raw data 2. Aggregated data 0-12hrs 3. Aggregated data 12-24hrs | X | |
| Time matched PK<br>Concentration for<br>urinary tetranor data<br>for tPGDM and<br>tPGEM | For each PD marker interval, use the upper bound as target time; e.g. for 0-2hr interval, 2hr is the target time Identify PK concentration with nominal time at the target time; If there is no PK sample taken at target time, use the PK concentration data with nominal time before but closest to target time; Use 0 PK concentration for placebo | X | X |
| Ratio of tPGDM/tPGEM # | Time matched ratio for tPGDM/tPGEM Three versions of data to be considered: 1.Creatinine corrected raw data 2. Creatinine corrected aggregated data 0-12hrs 3. Creatinine corrected aggregated data 12-24hrs 4. Aggregated data 24-48hrs | X | X |

# Urine tetranor and urine creatinine data should be considered as mass (Mass=Concentration\*Volume).

Raw data – Mass data for each of the intervals 0-2, 2-4, 4-6, 6-8, 8-12 &12-24. (predose and postdose)

Aggregated data 0-12hrs - Add the mass from each interval till 12 hrs (predose and postdose)

Aggregated data 12-24hrs - Mass from 12-24hr interval (predose and postdose)

Aggregated data 124-48hrs - Mass from 24-48hr interval (postdose)

### 10.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions

#### 10.1.2. Summary Measure

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 13.5.3. Reporting Standards for Pharmacokinetic)

#### 10.1.3. Population of Interest

The exploratory pharmacodynamics (and / or biomarker) analyses will be based on the PD population, unless otherwise specified.

## 10.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 10.1.4.1. Statistical Methodology Specification

#### 10.1.4.1.1. Statistical Methodology Specification for Part A (Single Dose)

#### Pharmacodynamic Statistical Analyses – Mixed Effect Model – Single Dose (Part A)

#### **Endpoint / Variables**

tPGDM, tPGEM, Creatinine, Creatinine corrected tPGDM and Creatinine corrected tPGEM (Aggregated values for predose 24-12hr & 12-0hr and postdose 0-12 hr, 12-24 hr & 24-48 hr)

#### **Model Specification**

Loge transformed values of the endpoints will be statistically analyzed using Mixed Model (MM).

- Fixed effect: dose, timepoint, dose\*timepoint
- Random effect: Subject

An unstructured covariance structure for the G matrix will be used.

- If this model fails to converge, alternative covariance structures may be considered.
- Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.

Analyses will be done with the MIXED Procedure in SAS, using the Kenward-Roger option to estimate denominator degrees of freedom and standard errors

#### **Model Checking & Diagnostics**

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted

#### Pharmacodynamic Statistical Analyses – Mixed Effect Model – Single Dose (Part A)

values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold.

#### Model Results Presentation

LS Geometric means and 90% CI are estimated for each dose as well as the estimate (90% CI) of change from baseline for each timepoint, using the time matched baseline.

Note: For post dose 24-48hrs baseline (predse) is not available

#### 10.1.4.1.2. Statistical Methodology Specification for Part B (Repeat Dose)

# Pharmacodynamic Statistical Analyses – Mixed Effect Model – Repeat Dose (Part B) Endpoint / Variables

tPGDM, tPGEM, Creatinine, Creatinine corrected tPGDM and Creatinine corrected tPGEM (Aggregated values for predose 24-12hr & 12-0hr and postdose 0-12 hr, 12-24 hr & 24-48 hr)

## **Model Specification**

Loge transformed values of the endpoints will be statistically analyzed using Mixed Model (MM).

- Fixed effect: timepoint, dose, timepoint\*dose
- Random effect: Subject

An unstructured covariance structure for the G matrix will be used.

- If this model fails to converge, alternative covariance structures may be considered.
- Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.

Analyses will be done with the MIXED Procedure in SAS, using the Kenward-Roger option to estimate denominator degrees of freedom and standard errors

### Model Checking & Diagnostics

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold.

#### **Model Results Presentation**

LS Geometric means and 90% CI are estimated for each dose as well as the estimate (90% CI) of change from baseline for each timepoint, using the time matched baseline.

Note: For post dose 24-48hrs baseline (predose) is not available

Consider Day -1(predose), Day1, Day 7, Day 10, Day 17

# 11. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

A detailed population PK/PD data analysis plan will be prepared in a separate RAP.

# 12. REFERENCES

GlaxoSmithKline Document Number 2018N361438\_03: Study Protocol of 209275, A Three-Part FTIH Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Repeat Oral Doses of GSK3439171A, in a Randomized, Double-Blind (sponsor unblinded), Placebo Controlled, Dose Escalation study and to Evaluate the Effect of Food on a Single Oral Dose of GSK3439171A in Healthy Adult Participants

# 13. APPENDICES

# 13.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

As Per Protocol Population is not defined, this section is not applicable.

# 13.2. Appendix 2: Schedule of Activities

# 13.2.1. Protocol Defined Schedule of Events

# SoA – Part A

| Part A- Single Dose | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Treatment Period [Days] (for each dosing period) | | | | | | Follow- | Notes<br>E.D = early | |
| Procedure | (up to 30<br>days<br>before Day<br>1) | -2 | -1 | 1 | 2 | 3 | 4 | E.D. | up<br>(~14±1<br>days<br>post last<br>dose) | discontinuation/withdrawal |
| Informed consent | Χ | | | | | | | | | |
| Inclusion and exclusion criteria (including drug screens) | X | | | X | | | | | | Recheck clinical status before randomization and/or 1st dose of study medication. |
| Demography | Χ | | | | | | | | | |
| Physical examination including height and weight | F | В | | | | | В | (B) | F | F: Full exam; B: Brief Exam; height is only taken once at screening |
| Part A- Single | e Dose | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| 1 | Screening | Treatment F | Period [Days] (fo | or each dosing perio | od) | | | | Follow-<br>up | Notes<br>E.D = early |
| Procedure | (up to 30<br>days<br>before Day<br>1) | -2 | -1 | 1 | 2 | 3 | 4 | E.D. | (~14±1<br>days<br>post last<br>dose) | discontinuation/withdrawal |
| Medical history (includes substance usage and family history of premature cardiovascular (CV) disease and any changes in health status occurring between screening and admission to the unit) | X | X | | | | | | | | Substances: Drugs, Alcohol, tobacco, and caffeine |
| Past and current medical conditions | Х | Х | | | | | | | | |
| Human<br>Immunodeficiency<br>Virus (HIV), Hepatitis<br>B and C screening | Х | | | | | | | | | If test otherwise performed within 3 months prior to first dose of study intervention, testing at screening is not required |
| Admission to Clinical Unit | | Х | | | | | | | | |
| Safety Laboratory<br>assessments<br>(include liver<br>chemistries) | X | Х | | Х | X | X | X | (X) | Х | Predose; 8 hr, 24 hr, and, 48 hr, and 72 hr post-dose and at follow-up visit |
| Routine Urinalysis | Х | | | Х | Х | Х | Х | (X) | Х | Predose; 8 hr, 24 hr, 48 hr, and 72 hr post-dose and at follow-up visit |

| Part A- Single | e Dose | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| - | Screening (up to 30 | | | or each dosing perio | | | I | | Follow-<br>up | Notes<br>E.D = early |
| Procedure | days<br>before Day<br>1) | -2 | -1 | 1 | 2 | 3 | 4 | E.D. | (~14±1<br>days<br>post last<br>dose) | discontinuation/withdrawal |
| 12-lead<br>Electrocardiogram<br>(ECG) | X | х | | <b>←</b> ====== | ) | (========= | <b>-</b> | (X) | Х | ECGs assessed at screening (triplicate) and admission (single). During treatment period ECGs assessed predose (triplicate at least 5 minutes (min) intervals) and single measurements postdose every 30 min for 1 hr, hourly up to 6 hr, and at 12 hr, 24 hr, 36 hr and 48 hr and 72 hr post-dose |
| Vital signs (pulse rate, blood pressure (bp), respiratory rate, and oral temperature) | X | х | | <b>←</b> ====== | :=====X | | ==== <b>-&gt;</b> | (X) | Х | Vitals assessed at screening (triplicate measurements for pulse and (bp)) (and admission (single measurements). During treatment period vitals assessed predose (triplicate measurements for pulse and bp) and postdose (single measurements) every 15 min for 1 hr, hourly up to 6 hr, then at 12 hr, 24 hr, 36 hr, 48 hr, and 72 hr postdose. |
| | | | | | | | | | | See Section 8.2.2 for further information |
| Randomization | | | | Х | | | | | | Randomization will occur before first dose in period 1. |

| Part A- Sing | le Dose | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Treatment F | Period [Days] (f | or each dosing perio | od) | | | | Follow- | Notes<br>E.D = early |
| Procedure | (up to 30<br>days<br>before Day<br>1) | -2 | -1 | 1 | 2 | 3 | 4 | E.D. | up<br>(~14±1<br>days<br>post last<br>dose) | discontinuation/withdrawal |
| Genetic sample | | | | X | | | | | | Any time predose on Day 1. This research may be described in a separate Informed Consent Form (ICF) or as part of a combined ICF. A separate signature is required where participant participation is optional |
| Study intervention | | | | Х | | | | | | |
| Telemetry | | | | X | | | | | | Telemetry performed starting 30 min ( $\pm 10$ min) pre-dose to 12 hr ( $\pm 20$ min) post-dose |
| Adverse Event (AE) review | | | | <b>←====</b> = | | =X======= | | (X) | Х | |
| Serious Adverse<br>Event (SAE) review | Х | | <b>←=====</b> | | =X====== | | :==→ | (X) | Х | |
| Concomitant medication review | Х | | <b>←===</b> | | ====X====== | <del>-</del> | | (X) | Х | |

| Part A- Singl | le Dose | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| 1 | Screening | Treatment F | Period [Days] (fo | or each dosing perio | od) | | | | Follow- | Notes<br>E.D = early |
| Procedure | (up to 30<br>days<br>before Day<br>1) | -2 | -1 | 1 | 2 | 3 | 4 | E.D. | up<br>(~14±1<br>days<br>post last<br>dose) | discontinuation/withdrawal |
| 24hr urine sampling | | | | | | | | | | <sup>1</sup> combined void for windows of 24-<br>22 hr, 22-20 hr, 20-18 hr, 18-16 hr,<br>16-12 hr, and 12-0 hr predose. |
| for Pharmacodynamics (PD) | | | X <sup>1</sup> | X <sup>2</sup> | X <sup>3</sup> | <b>X</b> <sup>3</sup> | | (X) | | <sup>2</sup> combined void for windows of 0-2<br>hr, 2-4 hr, 4-6 hr, 6-8 hr 8-12 hr,<br>and 12-24 hr post-dose<br><sup>3</sup> combined void for 24 hr |
| Blood sampling for<br>Pharmacokinetics<br>(PK) | | | | <b>←====</b> | X | | | (X) | | Predose, 5min, 30min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 18 hr, 24 hr, 36 hr, and 48 hr, 60 hr, and 72 hr post-dose |
| 24 hr Holter<br>Monitoring | | | | Х | | | | | | Predose through 24 hr post-dose |
| Discharge from<br>Clinical Unit | | | | | | | Х | (X) | | |

## **CONFIDENTIAL**

209275

The timing and number of planned study assessments, including safety, PK, PD/biomarker or other assessments may be altered during the course of the study based on newly available data (e.g., to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.

Any changes in the timing or addition of time points for any planned study assessments as the result of emerging pharmacokinetic/pharmacodynamic data from this study must be documented and approved by the relevant study team member and then archived in the sponsor and site study files, but will not constitute a protocol amendment. The Competent Authority (CA) and ethics committee (EC) will be informed of any safety issues that constitute a substantial amendment and require alteration of the safety monitoring scheme or amendment of the ICF. The changes will be approved by the CA and the EC before implementation.

## SoA – Part B

| | Screening | | | | | | | Inter | ventic | n Period | [Days] (f | or each d | osing co | hort) | | | | | E.D | Follow-<br>up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | (up to 30<br>days<br>before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5-7 | 8 | 9-11 | 12 | 13-14 | 15 | 16 | 17 | 18 | 19 | 20 | | (~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawal |
| Informed consent | Х | | | | | | | | | | | | | | | | | | | | |
| Inclusion and<br>exclusion criteria<br>(including drug<br>screens) | Х | Х | | | | | | | | | | | | | | | | | | | Recheck clinical status<br>before randomization and<br>prior to muscle biopsy/or<br>1st dose of study<br>medication. |
| Demography | Х | | | | | | | | | | | | | | | | | | | | |
| Full physical examination including height and weight | F | В | | | | | | | | | | | | | | | | В | (B) | F | F: Full exam; B: Brief<br>exam; height is only taken<br>once at screening |
| Medical history<br>(includes<br>substance usage<br>and family history<br>of premature CV<br>disease and any<br>changes in health<br>status occurring<br>between screening<br>and admission to<br>the unit) | х | х | | | | | | | | | | | | | | | | | | | Substances: Drugs,<br>Alcohol, tobacco, and<br>caffeine |

| Part B – Repeat Dos | ie . | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | | | | | | | Inter | /entic | n Period | [Days] (f | or each d | osing co | hort) | | | | | E.D | Follow-<br>up | |
| Procedure | (up to 30<br>days<br>before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5-7 | 8 | 9-11 | 12 | 13-14 | 15 | 16 | 17 | 18 | 19 | 20 | | (~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawal |
| Past and current medical conditions | Х | X | | | | | | | | | | | | | | | | | | | |
| HIV, Hepatitis B and C screening | Х | | | | | | | | | | | | | | | | | | | | If test otherwise<br>performed within 3<br>months prior to first dose<br>of study intervention,<br>testing at screening is not<br>required |
| Admission to<br>Clinical Unit | | Х | | | | | | | | | | | | | | | | | | | |
| Safety Laboratory<br>assessments<br>(include liver<br>chemistries) | х | | X | | | X | | X <sup>1</sup> | | X <sup>1</sup> | | | | | X <sup>1</sup> | | | Х | (X) | X <sup>1</sup> | Pre-randomization assessments for eligibility must be performed PRIOR to predose muscle biopsy Predose, 24 hr, and 48, and 72 hr post-Day 1 dose; additional timepoints may be added based on findings in Part A |
| | | | | | | | | | | | | | | | | | | | | | <sup>1</sup> Days 7, 11, 17, 20, and follow-up |

| | Screening | | | | | | | Inter | ventio | n Period | [Days] (t | or each d | osing co | hort) | | | | | E.D | Follow-<br>up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | (up to 30<br>days<br>before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5-7 | 8 | 9-11 | 12 | 13-14 | 15 | 16 | 17 | 18 | 19 | 20 | | (~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawal |
| Routine urinalysis | Х | Х | | | | x | | X <sup>2</sup> | | X <sup>2</sup> | | | | | X <sup>2</sup> | | | X <sup>2</sup> | (X) | X <sup>2</sup> | Predose, 24 hr, 48 hr, and 72 hr post-Day 1 dose; additional timepoints may be added based on findings in Part A <sup>2</sup> Days 7, 11,17, 20, and follow-up |

| Part B – Repeat Do | se | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | | | | | | | Inter | ventic | n Period | [Days] (f | or each d | losing co | hort) | | | | | E.D | Follow-<br>up | |
| Procedure | (up to 30<br>days<br>before<br>Day 1) | -2 | <b>–</b> 1 | 1 | 2 | 3 | 4 | 5-7 | 8 | 9-11 | 12 | 13-14 | 15 | 16 | 17 | 18 | 19 | 20 | | (~14±1<br>days<br>post<br>last<br>dose) | Notes E.D = early discontinuation/withdrawal |
| | | | | | | | | | | | | | | | | | | | | | Samples to be taken at midnight and 9am (±10 min) on Days -1 and 17 |
| | | | | | | | | | | | | | | | | | | | | | Samples taken at midnight<br>will be analysed for<br>adrenocorticotropic<br>hormone (ACTH) and<br>cortisol |
| Hormone<br>monitoring | | | X | | | | | | | | | | | | X | | | | (X) | | Samples taken at 9am will<br>be analysed for ACTH,<br>cortisol, luteinizing<br>hormone (LH), follicle<br>stimulating hormone<br>(FSH), thyroid stimulating<br>hormone (TSH), total<br>testosterone,<br>dihydrotestosterone (DHT),<br>triiodothyronine (T3), and<br>free thyroxine (free T4) |
| | | | | | | | | | | | | | | | | | | | | | See Section 8.2.7. in<br>Protocol for information<br>regarding monitoring of<br>abnormal hormone results |

| | | | | | | | | Inton | vont: | n Dorica | [Dove1 /f | or oach d | ooina co | hort) | | | | | E.D | Follow- | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening<br>(up to 30<br>days<br>before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5-7 | 8 | 9-11 | 12 | 13-14 | 15 | 16 | 17 | 18 | 19 | 20 | E.D | up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawal |
| 12-lead ECG | X | × | | <b>←</b> : | ==== | X <sup>5</sup> ==== | → | <b>X</b> 5 | | <b>X</b> ⁵ | | | <b>X</b> 5 | | <b>X</b> 5 | | | X⁵ | (X) | X | ECGs assessed at screening (triplicate measure) and admission (single measure). During treatment period ECGs assessed predose (triplicate measure at at least 5 min intervals) and post-dose (single measure) every 30 min for 1 hr, hourly up to 6 hr, at 12 hr post-dose then at 24 hr, 36 hr, 48 hr, and 72 hr post-dose |

| Part B – Repeat Dos | e | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | | | | | | | Inter | ventio | on Period | [Days] (f | or each d | osing co | hort) | | | | | E.D | Follow-<br>up | |
| Procedure | (up to 30<br>days<br>before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5-7 | 8 | 9-11 | 12 | 13-14 | 15 | 16 | 17 | 18 | 19 | 20 | | (~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawal |
| Vital signs (pulse rate, bp, respiratory rate, and oral temperature) | X | X | | | | X <sup>6</sup> | | | | | <b>X</b> <sup>7</sup> | | | | | > | (6 | | (X) | X | <sup>6</sup> Vitals assessed at screening (triplicate measurements for pulse and bp) and admission (single measurements). During treatment period vitals assessed predose (triplicate measurements for pulse and bp) and postdose (single measurements) every 15 min for 1 hr, hourly up to 6 hr, and at 12 hr, 24 hr, 36 hr, 48 hr, and 72 hr postdose <sup>7</sup> Vitals assessed once every 24 hr See Section 8.2.2. in Protocol for further information |
| Randomization | | | | Χ | | | | | | | | | | | | | | | | | |

| Part B – Repeat Dos | se | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | | | | | | | Inter | ventio | n Period | [Days] (t | for each d | osing co | hort) | | | | | E.D | Follow-<br>up | |
| Procedure | (up to 30<br>days<br>before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5-7 | 8 | 9-11 | 12 | 13-14 | 15 | 16 | 17 | 18 | 19 | 20 | | (~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawal |
| Genetic sample | | | | Х | | | | | | | | | | | | | | | | | Any time predose on Day 1 This research may be described in a separate ICF or as part of a combined ICF. A separate signature is required where participant participation is optional |
| Study intervention | | | | х | | | <b>←</b> = | | ==== | ====== | ===X=== | ====== | | | =→ | | | | | | |
| Telemetry | | | | х | | | | | | | | | | | | | | | | | Telemetry performed starting 30 (±10 min) predose to 12 hr (±20 min) post-dose |
| AE review | | | | | | | | <b>←</b> | ==== | ====== | ===== | | X | ==== | ===== | ==== | ==== | ==== | <i>&gt;</i> | | |
| SAE review | | | | | <b>←==</b> = | | ===== | | ==== | ===== | ===== | ====X== | | | ===== | | | | | <b>=</b> → | |
| Concomitant medication review | | | | | <b>←==</b> = | ===== | ===== | ===== | ==== | ====== | ===== | ====X== | ===== | ===== | ===== | ==== | ==== | ==== | ===== | <b>≔</b> → | |

| Part B – Repeat Dos | <u> </u> | | | | | | | 1.1 | | Б : . | 'D 1" | . , , | | 1 () | | | | | | Follow- | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening<br>(up to 30<br>days<br>before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5-7 | 8 | 9-11 | 12 | 13-14 | 15 | 16 | 17 | 18 | 19 | 20 | E.D | up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes E.D = early discontinuation/withdrawal |
| Urine sampling PD | | | X8 | X <sub>9</sub> | X9 | | | | | X <sup>9, 10</sup> | | | | | X9 | | | | (X) | | <sup>8</sup> combined void for windows of 24-22 hr, 22-20 hr, 20-18 hr, 18-16 hr, 16-12 hr, and 12-0 hr predose. <sup>9</sup> combined void for windows of 0-2 hr, 2-4 hr, 4-6 hr, 6-8 hr, 8-12 hr, and 12-24 hr post-dose <sup>10</sup> Day 10 only Aliquots will be removed prior to pooling for urine PK. Total urine volume will be recorded before aliquots for PD are removed. |

| | Screening | | | | | | | Inter | ventic | n Period | [Days] (f | or each d | osing co | hort) | | | | | E.D | Follow- | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | (up to 30<br>days<br>before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5-7 | 8 | 9-11 | 12 | 13-14 | 15 | 16 | 17 | 18 | 19 | 20 | | up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawa |
| 24h urine sampling<br>for PK and<br>metabolite profiling | | | x | X | х | | | | | | | | | | x | | | | (X) | | Voids from urine pharmacodynamic (PD) sampling windows will be combined into 0-24 hr pools on Day -1,1, and 17 after aliquoting for PD. These voids will be combined for PK/metabolite analysis only after aliquots for urine PD are removed See study reference manual (SRM) for details on samples and |

| Part B – Repeat Dos | se | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | | | | | | | Inter | ventic | n Period | [Days] (f | or each d | osing co | hort) | | | | | E.D | Follow-<br>up | |
| Procedure | (up to 30<br>days<br>before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5-7 | 8 | 9-11 | 12 | 13-14 | 15 | 16 | 17 | 18 | 19 | 20 | | (~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawal |
| Blood sampling for PK | | | | | ) | <b>(</b> 11 | | X <sup>12</sup> | | X <sup>12</sup> | | | X | 2 | | X | 11 | | (X) | | 11Day 1 and Day 17: Predose, 5 min, 30 min, 1 hr, 1. 5hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 18 hr, 24 hr, 36 hr, 48 hr, 60 hr, and 72 hr post-dose 12pre-dose samples collected on days 6,7, 9- 11 and 15-16 |
| Blood sampling for metabolite profiling | | | | | | X | | | | | | | | | | > | ( | | | | Day 1 and Day 17: Predose, 5 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 10 hr, 12 hr, 18 hr, 24 hr, 36 hr, 48 hr, 60 hr, and 72 hr post-dose |
| Blood sampling for<br>Pharmacodynamics<br>and biomarkers | | | | X <sup>13</sup> | X <sup>13</sup> | | | | | X <sup>14</sup> | | | | | X <sup>14</sup> | | | | (X) | | <sup>13</sup> Predose and 24 hr post-<br>dose on Day 1<br><sup>14</sup> Predose Days 10 and<br>17 |

| Part B – Repeat Do | se | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | | | | | | | Inter | ventic | n Period | [Days] (f | for each d | losing co | hort) | | | | | E.D | Follow-<br>up | |
| Procedure | (up to 30<br>days<br>before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5-7 | 8 | 9-11 | 12 | 13-14 | 15 | 16 | 17 | 18 | 19 | 20 | | (~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawal |
| | | | | | | | | | | | | | | | | | | | | | Muscle biopsies must be<br>performed AFTER clinical<br>safety assessments on<br>the corresponding days |
| Muscle Biopsy | | | X <sup>15</sup> | | | | | | | | | | | | X <sup>16</sup> | | | | (X) | | <sup>15</sup> Day -1 muscle biopsy to occur 1-6 hr after estimated timing of initial dose on Day 1. Time of sample collection to be recorded |
| ,,, | | | | | | | | | | | | | | | | | | | ( ) | | <sup>16</sup> Muscle Biopsy<br>performed any time during<br>pre-dose period; Day 17<br>muscle biopsy to occur<br>within 1-6 hr after last<br>dose administered |
| | | | | | | | | | | | | | | | | | | | | | Time of sample collection<br>to be recorded. Muscle<br>biopsy can be performed<br>at any time during pre-<br>dose period. |

| Part B – Repeat Dos | se | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening<br>(up to 30<br>days<br>before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | Interv | ventice 8 | on Period<br>9-11 | [Days] (f | or each d | osing co | hort) | 17 | 18 | 19 | 20 | E.D | Follow-up (~14±1 days post last dose) | Notes<br>E.D = early<br>discontinuation/withdrawal |
| Enterotest (bile sample collection) | | | | | | | | | | | | | | | Х | | | | | | For second or third dose-<br>level only (depending on<br>PK results in Part A) Enterotest capsule to be<br>swallowed ~2 hr after<br>dosing and removed ~7 hr<br>after dosing (~1 hr after<br>food cue) |
| Enterotest food cue | | | | | | | | | | | | | | | X | | | | | | For second or third dose-<br>level only (depending on<br>PK results in Part A) Food cue will be given 6<br>hr post-dose |
| Discharge from<br>Clinical Unit | | | | | | | | | | | | | | | | | | Х | (X) | | |

- The time to start the second dose in Part B can be modified based on the estimates of half-life from Part A.
- Duration of dosing in Part B can be modified based on the estimates of half-life from Part A.

## **CONFIDENTIAL**

209275

• The timing and number of planned study assessments, including safety, PK, PD/biomarker or other assessments may be altered during the course of the study based on newly available data (e.g., to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.

Any changes in the timing or addition of time points for any planned study assessments as the result of emerging pharmacokinetic/pharmacodynamic data from this study must be documented and approved by the relevant study team member and then archived in the sponsor and site study files, but will not constitute a protocol amendment. The CA and EC will be informed of any safety issues that constitute a substantial amendment and require alteration of the safety monitoring scheme or amendment of the ICF. The changes will be approved by the CA and the EC before implementation.

| Part B .2- 7 Day Rep | eat Dose | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screenin<br>g<br>(up to 30<br>days<br>before<br>Day 1) | | | | | | Int | erveni | tion Peri | od [Days] | (for eacl | n dosing co | ohort) | | | | E.D | Follow-<br>up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawa<br>I |
| | Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | | | |
| Informed consent | Х | | | | | | | | | | | | | | | | | | |
| Inclusion and exclusion criteria (including drug screens) | X | Х | | | | | | | | | | | | | | | | | Recheck clinical status<br>before randomization and<br>prior to muscle biopsy/or<br>1st dose of study<br>medication. |
| Demography | Х | | | | | | | | | | | | | | | | | | |
| Full physical examination including height and weight | F | В | | | | | | | | | | | | | | В | (B) | F | F: Full exam; B: Brief<br>exam; height is only taken<br>once at screening |
| Medical history (includes substance usage and family history of premature CV disease and any changes in health status occurring between screening and admission to the unit) | X | Х | | | | | | | | | | | | | | | | | Substances: Drugs,<br>Alcohol, tobacco, and<br>caffeine |

| Part B .2- 7 Day Re | peat Dose | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screenin<br>g<br>(up to 30<br>days<br>before | | | | | | Inte | erven | tion Peri | od [Days] | (for eacl | n dosing co | ohort) | | | | E.D | Follow-<br>up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawa |
| | Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | | | |
| Past and current medical conditions | Х | Х | | | | | | | | | | | | | | | | | |
| HIV, Hepatitis B and C screening | X | | | | | | | | | | | | | | | | | | If test otherwise<br>performed within 3<br>months prior to first dose<br>of study intervention,<br>testing at screening is not<br>required |
| Admission to<br>Clinical Unit | | Х | | | | | | | | | | | | | | | | | |
| Safety Laboratory<br>assessments<br>(include liver<br>chemistries) | X | | X | | | x | | | | X <sup>1</sup> | | | X1 | | | X <sup>1</sup> | (X) | X1 | Pre-randomization assessments for eligibility must be performed PRIOR to predose muscle biopsy Predose, 24 hr, and 48, and 72 hr post-Day 1 dose; additional timepoints may be added based on findings in Part A ¹Days 7, 10, 13, and follow-up |

| Procedure | Screenin<br>g<br>(up to 30<br>days<br>before<br>Day 1) | | | | | | Int | tervent | tion Peri | od [Days] | (for each | n dosing c | ohort) | | | | E.D | Follow-<br>up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawa |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | | , | |
| Routine urinalysis | Х | X | | | | X | | | | X <sup>2</sup> | | | X <sup>2</sup> | | | X <sup>2</sup> | (X) | X <sup>2</sup> | Predose, 24 hr, 48 hr,<br>and 72 hr post-Day 1<br>dose; additional<br>timepoints may be added<br>based on findings in Part<br>A<br><sup>2</sup> Days 7, 10, 13, and<br>follow-up |

| Part B .2- 7 Day Rep | peat Dose | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screenin<br>g<br>(up to 30<br>days<br>before<br>Day 1) | | | | | | Inte | erveni | tion Peri | od [Days] | (for eacl | n dosing co | ohort) | | | | E.D | Follow-<br>up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawa<br>I |
| | Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | | | |
| | | | | | | | | | | | | | | | | | | | Samples to be taken at midnight and 9am (±10 min) on Days -1 and 10 |
| | | | | | | | | | | | | | | | | | | | Samples taken at midnight<br>will be analysed for<br>adrenocorticotropic<br>hormone (ACTH) and<br>cortisol |
| Hormone<br>monitoring | | | X | | | | | | | | | | X | | | | | | Samples taken at 9am will be analysed for ACTH, cortisol, luteinizing hormone (LH), follicle stimulating hormone (FSH), thyroid stimulating hormone (TSH), total testosterone, dihydrotestosterone (DHT), triiodothyronine (T3), and free thyroxine (free T4) |
| | | | | | | | | | | | | | | | | | | | See Section 8.2.7. in<br>Protocol for information<br>regarding monitoring of<br>abnormal hormone results |

| Part B .2- 7 Day Rep | peat Dose | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screenin<br>g<br>(up to 30<br>days<br>before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | Int | erven | tion Perio | od [Days] | (for each | n dosing co | ohort) | 11 | 12 | 13 | E.D | Follow-<br>up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawa<br>I |
| 12-lead ECG | X | X | | | <b>-</b> | | | | | X <sup>5</sup> | | | X <sup>5</sup> | | | X <sup>5</sup> | (X) | X5 | ECGs assessed at screening (triplicate measure) and admission (single measure). During treatment period ECGs assessed predose (triplicate measure at at least 5 min intervals) and post-dose (single measure) every 30 min for 1 hr, hourly up to 6 hr, at 12 hr post-dose then at 24 hr, 36 hr, 48 hr, and 72 hr post-dose |
| | | | | | | | | | | | | | | | | | | | <sup>5</sup> Days 7,10, 13, and<br>Follow-up Post-dose at<br>Cmax based on observed<br>Cmax in Part A (currently<br>estimated to occur at ~2<br>hr post dose), except for<br>Day 13. Day 13 ECG to<br>occur any time before<br>Discharge |

| Part B .2- 7 Day Rep | eat Dose | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screenin<br>g<br>(up to 30<br>days<br>before<br>Day 1) | -2 | -1 | 1 | 2 | 3 | Int | ervent | tion Perio | od [Days] | (for each | n dosing c | ohort) | 11 | 12 | 13 | E.D | Follow-<br>up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawa<br>I |
| Vital signs (pulse rate, bp, respiratory rate, and oral temperature) | X | x | | | | <b>X</b> 6 | | | | | | <b>X</b> <sup>7</sup> | | | | X6 | (X) | X | 6Vitals assessed at screening (triplicate measurements for pulse and bp) and admission (single measurements). During treatment period vitals assessed predose (triplicate measurements for pulse and bp) and postdose (single measurements) every 15 min for 1 hr, hourly up to 6 hr, and at 12 hr, 24 hr, 36 hr, 48 hr, and 72 hr post-dose 7Vitals assessed once every 24 hr See Section 8.2.2. in Protocol for further information |
| Randomization | | | | Х | | | | | | | | | | | | | | | |

| Part B .2- 7 Day Rep | peat Dose | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screenin<br>g<br>(up to 30<br>days<br>before<br>Day 1) | | | | | I | Int | 1 | 1 | · | | n dosing c | ·<br>T | | | | E.D | Follow-<br>up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes E.D = early discontinuation/withdrawa |
| | | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | | | |
| Genetic sample Study intervention | | | | x | | | <b>←===</b> | | | X | | | <b>-</b> | | | | | | Any time predose on Day 1 This research may be described in a separate ICF or as part of a combined ICF. A separate signature is required where participant participation is optional |
| Telemetry | | | | х | | | | | | | | | | | | | | | Telemetry performed starting 30 (±10 min) predose to 12 hr (±20 min) post-dose |
| AE review | | | | + | -=== | | | | | ===== | | X===== | ====== | ===== | ===== | | | ===> | |
| SAE review | <b>←====</b> | ==== | ===== | ===== | ===== | ===== | ====== | | :===== | ==X==== | ===== | ====== | ====== | ===== | ===== | | ======= | ====→ | |
| Concomitant medication review | <b>←===</b> | ==== | ===== | ==== | ==== | ===== | ===== | ==== | ===== | ====== | -X==== | :===== | ===== | ===== | ===== | ===== | ====== | ==→ | |

| Part B .2- 7 Day Re | oeat Dose | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screenin<br>g<br>(up to 30<br>days<br>before | | | | | | Int | ervent | tion Perio | od [Days] | (for eacl | n dosing co | ohort) | | | | E.D | Follow-<br>up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawa<br>I |
| | Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | | , | |
| Urine sampling PD | | | X8 | × | 'œ' | | | | | Χ9 | | | X | 9 | | | (X) | | 8combined void for windows of 24-22 hr, 22-20 hr, 20-18 hr, 18-16 hr, 16-12 hr, and 12-0 hr predose. 9combined void for windows of 0-2 hr, 2-4 hr, 4-6 hr, 6-8 hr, 8-12 hr, and 12-24 hr post-dose Aliquots will be removed prior to pooling for urine PK. Total urine volume will be recorded before aliquots for PD are removed. |

| Part B .2- 7 Day Rep | peat Dose | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | before Day 1) | | | | Intervention Period [Days] (for each dosing cohort) | | | | | | | | | E.D | Follow-<br>up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawa<br>I | | |
| | Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | | |
| 24h urine sampling<br>for PK and<br>metabolite profiling | | | X | | X | | | | | | | | х | ( | | | (X) | Voids from urine pharmacodynamic (PD) sampling windows will be combined into 0-24 hr pools on Day -1,1, and 10 after aliquoting for PD. These voids will be combined for PK/metabolite analysis only after aliquots for urine PD are removed |
| | | | | | | | | | | | | | | | | | | See study reference<br>manual (SRM) for details<br>on samples and<br>processing |

| Part B .2- 7 Day Rep | peat Dose | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screenin<br>g<br>(up to 30<br>days<br>before<br>Day 1) | | | | Intervention Period [Days] (for each dosing cohort) | | | | | | | E.D | Follow-<br>up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawa<br>I | | | | |
| | Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | | |
| Blood sampling for PK | | | | | | X <sup>10</sup> | | | X <sup>11</sup> | X <sup>11</sup> | | X <sup>11</sup> | | Х | 10 | | (X) | 10Day 1 and Day 10:<br>Predose, 5 min, 30 min, 1<br>hr, 1. 5hr, 2 hr, 3 hr, 4 hr,<br>6 hr, 8 hr, 10 hr, 12 hr, 18<br>hr, 24 hr, 36 hr, 48 hr, 60<br>hr, and 72 hr post-dose |
| Blood sampling for metabolite profiling | | | | | | X | | | | | | | | > | ( | | | Day 1 and Day 10<br>Predose, 5 min, 30 min, 1<br>hr, 1.5 hr, 2 hr, 3 hr, 4 hr,<br>6 hr, 8 hr, 10 hr, 12 hr, 18<br>hr, 24 hr, 36 hr, 48 hr, 60<br>hr, and 72 hr post-dose |
| Blood sampling for<br>Pharmacodynamic<br>s and biomarkers | | | | X <sup>12</sup> | X <sup>12</sup> | | | | | X <sup>13</sup> | | | X <sup>13</sup> | | | | (X) | <sup>12</sup> Predose and 24 hr post-<br>dose on Day 1<br><sup>13</sup> Predose Days 7 and 10 |

| Part B .2– 7 Day Repeat Dose | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screenin<br>g<br>(up to 30<br>days<br>before<br>Day 1) | | | | Intervention Period [Days] (for each dosing cohort) | | | | | | E.D | Follow-<br>up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawa<br>I | | | | | |
| | | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | | |
| | | | | | | | | | | | | | | | | | | Muscle biopsies must be performed AFTER clinical safety assessments on the corresponding days |
| Muscle Biopsy | | | X <sup>14</sup> | | | | | | | | | | <b>X</b> <sup>15</sup> | | | | (X) | <sup>14</sup> Day -1 muscle biopsy to occur 1-6 hr after estimated timing of initial dose on Day 1. Time of sample collection to be recorded |
| | | | | | | | | | | | | | | | | | | <sup>15</sup> Day 10 muscle biopsy<br>to occur within 1-6 hr after<br>last dose administered |
| | | | | | | | | | | | | | | | | | | Time of sample collection<br>to be recorded. Muscle<br>biopsy can be performed<br>at any time during pre-<br>dose period. |

| Part B .2– 7 Day Re | Screenin<br>g<br>(up to 30<br>days<br>before | | | | Intervention Period [Days] (for each dosing cohort) | | | | | | | | | | E.D | Follow-<br>up<br>(~14±1<br>days<br>post<br>last<br>dose) | Notes<br>E.D = early<br>discontinuation/withdrawa | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day 1) | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | | , |
| Discharge from<br>Clinical Unit | | | | | | | | | | | | | | | | Х | (X) | |

- The time to start the second dose in Part B can be modified based on the estimates of half-life from Part A.
- Duration of dosing in Part B can be modified based on the estimates of half-life from Part A.
- The timing and number of planned study assessments, including safety, PK, PD/biomarker or other assessments may be altered during the course of the study based on newly available data (e.g., to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.
- Any changes in the timing or addition of time points for any planned study assessments as the result of emerging pharmacokinetic/pharmacodynamic data from this study must be documented and approved by the relevant study team member and then archived in the sponsor and site study files, but will not constitute a protocol amendment. The CA and EC will be informed of any safety issues that constitute a substantial amendment and require alteration of the safety monitoring scheme or amendment of the ICF. The changes will be approved by the CA and the EC before implementation.

| Part C- Food Effe | ct | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Treatment Period | Days] (with or without food | ) | | | | Follow-<br>up | |
| | Screening<br>(up to 30<br>days<br>before Day<br>1) | <u>-1</u> | 1 | 2 | 3 | 4 | E.D. | (~14±1<br>days<br>post<br>last<br>dose) | Notes E.D = early discontinuation/withdrawal |
| Informed consent | Х | | | | | | | | |
| Inclusion and<br>exclusion criteria<br>(including drug<br>screens) | Х | | Х | | | | | | Recheck clinical status<br>before randomization and/or<br>1st dose of study medication. |
| Demography | Х | | | | | | | | |
| Physical examination including height and weight | F | В | | | | В | (B) | F | F: Full exam; B: Brief Exam;<br>height is only taken once at<br>screening |

| Part C- Food Effe | ect | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| . Lit o i ood Ello | | Treatment Period | Days] (with or without food | ) | | | | Follow- | |
| | Screening<br>(up to 30<br>days<br>before Day<br>1) | <b>-1</b> | 1 | 2 | 3 | 4 | E.D. | up (~14±1 days post last dose) | Notes E.D = early discontinuation/withdrawal |
| Medical history (includes substance usage and family history of premature CV disease and any changes in health status occurring between screening and admission to the unit) | X | X | | | | | | | Substances: Drugs, Alcohol, tobacco, and caffeine |
| Past and current medical conditions | Х | Х | | | | | | | |
| HIV, Hepatitis B and C screening | х | | | | | | | | If test otherwise performed within 3 months prior to first dose of study intervention, testing at screening is not required |
| Admission to Clinical Unit | | Х | | | | | | | |

| Part C- Food Effe | ct | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Treatment Period | [Days] (with or without food) | ) | | | | Follow-<br>up | |
| | Screening<br>(up to 30<br>days<br>before Day | <b>-1</b> | 1 | 2 | 3 | 4 | E.D. | (~14±1<br>days<br>post<br>last<br>dose) | Notes E.D = early discontinuation/withdrawal |
| Safety<br>Laboratory<br>assessments<br>(including liver<br>chemistries) | Х | X | X | Х | Х | Х | (X) | Х | Predose; 8 hr, 24 hr, 48 hr,<br>and 72 hr post-dose and at<br>follow-up visit |
| Routine<br>Urinalysis | х | | X | Х | Х | X | (X) | X | Predose; 8 hr, 24 hr, 48 hr,<br>and 72hr post-dose and at<br>follow-up visit |
| 12-lead ECG | X | X | <b>←</b> ========== | :=====X====== | | <b>-</b> | (X) | Х | ECGs assessed at screening (triplicate) and admission (single). During treatment period ECGs assessed predose (triplicate at least 5 min intervals) and single measurements postdose every 30 min for 1 hr, hourly up to 6 hr, and at 12 hr, 24 hr, 36 hr, 48 hr, and 72 hr post-dose |

| Part C- Food Effe | ct | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Treatment Period [ | Days] (with or without food | | | Follow-<br>up | | | |
| | Screening<br>(up to 30<br>days<br>before Day<br>1) | -1 | 1 | 2 | 3 | 4 | E.D. | (~14±1<br>days<br>post<br>last<br>dose) | Notes E.D = early discontinuation/withdrawal |
| Vital signs (pulse rate, bp, respiratory rate, and oral temperature) | X | X | <b>←</b> ===== | X=: | | <b>&gt;</b> | (X) | X | Vitals assessed at screening (triplicate measurements for pulse and bp) and admission (single measurements). During treatment period vitals assessed predose (triplicate measurements for pulse and bp) and postdose (single measurements) every 15 min for 1 hr, hourly up to 6 hr, and at 12 hr, 24 hr, 36 hr, 48 hr, and 72 hr post-dose See Section 8.2.2. in Protocol for further information |
| Randomization | | | Х | | | | | | |

| Part C- Food Effe | ct | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Treatment Perio | d [Days] (with or without food | ) | | | | Follow-<br>up | |
| | Screening<br>(up to 30<br>days<br>before Day<br>1) | <b>-</b> 1 | 1 | 2 | 3 | 4 | E.D. | (~14±1<br>days<br>post<br>last<br>dose) | Notes E.D = early discontinuation/withdrawal |
| Genetic sample | | | X | | | | | | Sample can be obtained at any point during dosing. This research may be described in a separate ICF or as part of a combined ICF. A separate signature is required where participant participation is optional |
| Test Meal | | | X | | | | | | Fed Arm only. See Section<br>5.3.1. in Protocol for timings<br>regarding meals, fasting, and<br>treatment administration |
| Study intervention | | | Х | | | | | | |
| Telemetry | | | Х | | | | | | Telemetry performed starting 30 min (±10 min) pre-dose to 12hrs (±20 min) post-dose |
| AE review | | | <b>←==</b> : | X=- | -====== | <del></del> | (X) | Х | |
| SAE review | Х | | <del>(</del> | XX | | (X) | | | |

| Part C- Food Effe | ct | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Caraaning | Treatment Period | [Days] (with or without food | i) | | | | Follow-<br>up | |
| | Screening<br>(up to 30<br>days<br>before Day<br>1) | <b>-1</b> | 1 | 2 | 3 | 4 | E.D. | (~14±1<br>days<br>post<br>last<br>dose) | Notes E.D = early discontinuation/withdrawal |
| Concomitant medication review | х | <b>←==</b> | | XX | | ===→ | (X) | Х | |
| Blood sampling for PK | | | <b>←===</b> = | X- | ======================================= | =→ | (X) | | <sup>3</sup> Predose, 5 min, 30 min, 1<br>hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6<br>hr, 8 hr, 10 hr, 12 hr, 18 hr,<br>24 hr, 36 hr, and 48 hr, 60 hr,<br>and 72 hr post-dose |
| Discharge from<br>Clinical Unit | | | | | | Х | (X) | | |

- Duration of dosing in Part C can be modified based on the estimates of half-life from Part A.
- The timing and number of planned study assessments, including safety, PK, PD/biomarker or other assessments may be altered during the course of the study based on newly available data (e.g., to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.

Any changes in the timing or addition of time points for any planned study assessments as the result of emerging pharmacokinetic/pharmacodynamic data from this study must be documented and approved by the relevant study team member and then archived in the sponsor and site study files, but will not constitute a protocol amendment. The CA and EC will be informed of any safety issues that constitute a substantial amendment and require alteration of the safety monitoring scheme or amendment of the ICF. The changes will be approved by the CA and the EC before implementation.
# 13.3. Appendix 3: Assessment Windows

Nominal time will be used for all analysis except PK analysis where planned and actual time will be used.

# 13.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 13.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date + 3 days |
| Post-Treatment | Date > Study Treatment Stop Date + 3 days |

Note: Estimated half-life of GSK3439171 is approx. 13 hours. The maximum of (5 halflives  $\sim$  65 hours  $\sim$  3days) and after the Study Treatment End Date, lag time have been considered to be 3 days to define the end of treatment phase.

#### 13.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days, prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 13.5. Appendix 5: Data Display Standards & Handling Conventions

## 13.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : us1salx00259 |
| HARP Compound | : /arenv/arprod/gsk3439171/mid209275/final_01 |
| Analysis Datasets | |
| Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.0 | |
| Generation of RTF Files | |
| RTF files will be generated for SAC. | |

## 13.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.

• The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### Planned and Actual Time

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures. However, for baseline consideration if the latest predose is an unscheduled visit, then as per the baseline definition, this will be considered as baseline. And unscheduled visits will be taken into consideration for calculating worst-case post baseline value in ECG displays as well.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

#### 13.5.3. Reporting Standards for Pharmacokinetic

| <b>Concentration Data</b> | |
|---|---|
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Pharmacokinetic Parameters | |
| Descriptive | N, n, geometric mean, 90% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation |
| Summary Statistics | (CVb (%)) will be reported. |
| (Log Transformed) | |

| | CVb (%) = $\sqrt{(\exp(SD2) - 1) * 100}$ [NOTE: SD = SD of loge transformed data] |
|---|---|
| | Following steps can be used to calculate 90% CI for PK parameters: |
| | Standard Error = [(Geometric Stdev-1)/Sqrt(N)], |
| | Margin of Error = [Standard Error * 1.645], and |
| | $CI = [Geometric Mean \pm Margin of Error]$ |
| Parameters Not<br>Being Log | tmax, t½ |
| Transformed | |
| Summary Tables | Cmax, tmax, AUC(0-т), AUC(0-t), AUC (0-∞), AUC (Ro), |
| • | Rcmax, Ct, t1/2, Rss, Ae, fe, CLr, as data permit |
| Listings | Include PK Parameters Cmax, tmax, AUC(0-τ), AUC(0-t), AUC (0-∞), AUC (Ro), Rcmax, Cτ, t1/2, Rss, Ae, fe, CLr, as data |
| | Permit |
| Graphical Displays | |
| Refer to IDSL Statistical Principles 7.01 to 7.13 and Standards for the Transfer and | |
| Reporting of PK Data | Reporting of PK Data using HARP. |

| Pharmacokinetic Con | Pharmacokinetic Concentration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the noncompartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to [Insert document name]. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Para | Pharmacokinetic Parameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | The following PK parameters will be derived by the Programmer: [Insert PK parameters, e.g. C24, C12, AUC/Dose] |
| Pharmacokinetic Para | Pharmacokinetic Parameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | No. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. |

# 13.6. Appendix 6: Derived and Transformed Data

#### 13.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day and Period Study Day

In PART A and C, Period Study day is calculated as the number of days from first Dose

Date in the period for each subject as follows:

- Ref Date = Missing → Period Study Day = Missing
- Ref Date < First Dose Date in the period → Period Study Day = Ref Date First Dose Date in the period
- Ref Data ≥ First Dose Date in the period → Period Study Day = Ref Date First Dose Date in the period + 1

In Part A, B & C: Study day is calculated as the number of days from First Dose Date in each Cohort for each subject as:

- Ref Date = Missing → Study Day = Missing
- Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
- Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## Change from baseline and Percentage change from baseline definition

Change from Baseline = Post-Dose Visit Value – Baseline (For Part A & C, corresponding period baseline should be considered as baseline)

Percentage Change from Baseline = ((Post-Dose Visit Value – Baseline)/Baseline)\*100 (For Part A & C, corresponding period baseline should be considered as baseline)

- Unless otherwise specified, the baseline definitions specified in Section 5.2 Baseline Definition will be used for derivations for endpoints / parameters and indicated on summaries and listings
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing

#### **Displays**

- Compound ID should be used as GSK3439171 for the displays
- Listings: Since it is single site study, site id and investigator id will be included in 'Listing of Planned and Actual Treatment' and will be excluded from other Listings.
- Safety summaries and figures:
  - Part A and B, 'All treatment' total (Subjects on treatment except placebo) should be included and footnote to indicate this. Part C overall
    'Total' should be included.
  - o Part A and C, in Lab, Vitals and ECG displays, Day -2 and -1(if available) should be included for absolute value displays.
  - o Part B in Lab, Vitals and ECG displays, Day -2 and -1(if available) should be included for absolute value displays along with screening and follow up data. And for change from baseline and percentage change from baseline displays follow up data should be included

### 13.6.2. Study Population

#### **Treatment Compliance**

Treatment compliance will be calculated based on the formula:

### Treatment Compliance = Number of Actual Doses / (Planned Treatment Duration in Days \* Frequency)

• Frequency is 2 for BID and 1 for QD. Treatment compliance could be greater than 100% if there are events of overdose. Cumulative compliance (since Day 1) at each visit will be calculated.

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

#### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### Cumulative Dose = Sum of (Number of Days x Total Daily Dose)

If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

## 13.6.3. Safety

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01</li>
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1</li>

#### **ECG Parameters**

#### **RR Interval**

- If RR interval (msec) is not provided directly, then RR can be derived as:
  - [1] If QTcF is machine read, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

• If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value. THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the ClinBase, corrected QT intervals by Fredericia's (QTcF) formula will be calculated in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcF will be derived as:

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### 13.6.4. Pharmacokinetic

#### **PK Parameters**

The PK Population will include all subjects who undergo PK sampling and have evaluable PK assay results.

 See Table 2. Derived Pharmacokinetic Parameters (Primary end points) and Table 3. Derive d Pharmacokinetic Parameters (Secondary end points) for derived Pharmacokinetic parameters

# 13.7. Appendix 7: Reporting Standards for Missing Data

# 13.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as 'A participant is considered to have completed the study if he/she has completed all phases of the study including or the last scheduled procedure shown in the SoA.'</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 13.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 13.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse Events | The Clinbase allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used. |
| | <ul> <li>Completely missing start or end dates will remain missing, with no imputation<br/>applied. Consequently, time to onset and duration of such events will be<br/>missing.</li> </ul> |
| Concomitant<br>Medications/Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day</li> </ul> |

| Element | Reporting Detail |
|---|---|
| | (dependent on the month and year) and 'Dec' will be used for the month. |
| | The recorded partial date will be displayed in listings. |
| | For each period in crossover design: |
| | <ul> <li>If start date is completely missing, then we assume the medication</li> </ul> |
| | has been taken from the beginning of the study |
| | <ul> <li>If stop date is completely missing, then we assume the medication</li> </ul> |
| | has been taken until the end of the study |

# 13.7.2.2. Handling of PK Concentration Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument.</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all</li> </ul> |
| | <ul> <li>data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented |
| | along with the reason for exclusion in the clinical study report. |

# 13.7.2.3. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| Imputation | <ul> <li>No imputation will be performed for missing data</li> </ul> |

# 13.8. Appendix 8: Values of Potential Clinical Importance

# 13.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | Detic of | Male | | 0.54 |
| Hematocrit | Ratio of | Female | | 0.54 |
| | ' | $\Delta$ from BL | ↓0.075 | |
| | a/I | Male | | 180 |
| Haemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | $\Delta$ from BL | | <b>↑ 44.2</b> |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | .5 | 1.23 |
| Phosphorus | mmol/L | | .8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Creatine Kinase (CK) | | | | >500 U/I |
| Liver Function | | | | |
| Test Analyte | Units | Category | Clinical Concern Range | |
| ALT/SGPT | U/L | High | ≥ 2x | ULN |
| AST/SGOT | U/L | High | ≥ 2x | ULN |
| AlkPhos | U/L | High | ≥ 2x ULN | |
| T Bilirubin | µmol/L | High | ≥ 1.5x ULN | |
| | µmol/L | | 1.5xULN | Γ. Bilirubin |
| T. Bilirubin + ALT | | High | +<br>≥ 2x ULN ALT | |
| | U/L | | 27.01 | <b>.</b> |

# 13.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | >450 |
| Absolute PR Interval | msec | <110 | >220 |
| Absolute QRS Interval | msec | <75 | >110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | >60 |

# 13.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | <85 | >160 |
| Diastolic Blood Pressure | mmHg | <45 | >100 |
| Heart Rate | bpm | <40 | >110 |

# 13.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses

PopPK will be performed under a separate RAP and will be reported separately

# 13.10. Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses

A detailed population PK/PD data analysis plan will be prepared in a separate RAP.

# 13.11. Appendix 11: Abbreviations & Trade Marks

# 13.11.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | |
| | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| טטטר | Study Data Standardization Flan |

| Abbreviation | Description |
|--------------|------------------------------|
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| SR | Safety Review |

# 13.11.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| NONMEM |
| SAS |
| WinNonlin |

## 13.12. Appendix 12: List of Data Displays

- PROGRAMMING NOTES: Where applicable, programming notes can be included to supplement and/or highlight specific information to aid with display generation.
  - Consideration should be given to any changes to the standard GSK IDSL displays or inclusion of optional columns for safety reporting.
  - If applicable, provide additional information to aid generation of graphical displays (e.g. if a multiple panel plot is being generated then details such as the number of rows / columns, panel by variable, legend variable etc may be included).
  - Consideration should be given for additional level of instructions for any outsourced studies, so as to ensure clarity for generating each display to the expected specifications.
  - Note: Small studies (e.g. early phase studies) or where sample sizes or event rates are small, study teams may choose to omit certain summary tables where a listing of the data would be sufficient (See IDSL Principle 4.21 Minimal Analysis). The lead RAP author / RAP Team should consult and get agreement from medical writing / CSR writer that listings would be sufficient for the study.

## 13.12.1. Data Display Numbering

- NOTE: The numbering of data displays is now driven by best practices outlined for the
  development of the Clinical Study Report but the numbering scheme should be utilised
  for all reporting efforts. For listings utilise sequential numbering for ICH and Other
  Listings.
- <u>Automation:</u> Numbering of data displays is automated within tables. If rows are added or deleted, the numbering of displays will be automatically updated. Therefore, when updating sections based on the order of objectives / endpoints in the protocol, <u>rename</u> <u>section headings</u> rather than rearranging sections using cut and paste options.

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|-------------|-------------|
| Study Population | 1.1 to 1.33 | - |
| Safety | 3.1 to 3.67 | 3.1 to 3.28 |
| Pharmacokinetic | 4.1 to 4.26 | 4.1 to 4.15 |
| Pharmacodynamic and / or Biomarker | 6.1 to 6.9 | 6.1 to 6.16 |
| Section | Listi | ngs |
| ICH Listings | 1 to | 110 |
| Non-ICH Listings | 111 to | 134 |
| Other Listings | 13 | 35 |

#### 13.12.2. Mock Example Shell Referencing

• **Mock Example Shells:** Only to be provided if not covered by GSK IDSL, or if there are major changes to the standard data displays.

 Alternately, provide an appropriate GSK IDSL data standard reference and include details in the programming notes column for the display to be generated.

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Section 13.13: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|-----------------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic / Biomarker | PD_Fn | PD_Tn | PD_Ln |

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 13.12.3. Deliverables

- Delivery Priority: If applicable, can provide information on whether specific outputs are required at times other than statistical analysis complete (SAC) or to provide an order of displays to be generated so as to facilitate and manage reporting.
- Example where the deliverable priority may be used are:
  - Decision Critical Data Reporting: For example, this may include endpoints reported prior to SAC that are required for making critical decisions for the compound.
  - Partial Data Reporting: For example, this may include a study conducted in multiple parts where there will be unblinding and reporting of one or more parts of the study prior to database freeze.
  - Exploratory Data Reporting: For example, this may include endpoints that are
    potentially analysed post SAC (e.g. TAQMAN data). These may not be intended
    for the CPSR report and as such would not need to have a table or figure number.
  - Output for Presentation Purposes Only: For example, this may include combining output with data from other sources for presentation purposes. These would not be intended for the CPSR report and as such would not need to have a display number.

| Delivery [Priority] [1] | Description |
|---|---|
| SR | Safety Review (after completing Part A and Part B cohort 1& 2) |
| SAC | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 13.12.4. Study Population Tables

- The requirements for each display (i.e. IDSL, ICH etc.) specified in the programming notes may be retained, all other red reference notes should be deleted.
- Select appropriate standard based on study design (i.e. parallel vs cross-over), when applicable.
- The ADaM datasets for the Core Study Population/Safety displays can be found in the IDSL Library under Reference → Statistical Displays → ADaM Datasets for Core RAP Displays

| Study Po | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject [ | Disposition | | | | • |
| 1.1. | Safety | CP_ES1 | Summary of Subject Status and Reason for Study Withdrawal - Part A | by Cohort | SAC |
| 1.2. | Safety | CP_ES1 | Summary of Subject Status and Reason for Study Withdrawal - Part B | by Cohort | SAC |
| 1.3. | Safety | CP_ES1 | Summary of Subject Status and Reason for Study Withdrawal - Part C | By Cohort- since only one cohort,<br>'Total' column | SAC |
| 1.4. | Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment – Part B | By Dose | SAC |
| 1.5. | Safety | ES4 | Summary of Participant Disposition at Each Study Epoch - Part A | By Cohort | SAC |

| Study P | opulation Tab | les | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.6. | Safety | ES4 | Summary of Participant Disposition at Each Study Epoch - Part C | By Cohort | SAC |
| 1.7. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure - Part A | by Cohort | SAC |
| 1.8. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure - Part B | by Cohort | SAC |
| 1.9. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure - Part C | By Cohort- since only one cohort,<br>'Total' column | SAC |
| Protoco | Deviation | | | | |
| 1.10. | Safety | DV1 | Summary of Important Protocol Deviations - Part A | By dose | SAC |
| 1.11. | Safety | DV1 | Summary of Important Protocol Deviations - Part B | By Dose | SAC |
| 1.12. | Safety | DV1 | Summary of Important Protocol Deviations - Part C | By Dose | SAC |
| Populati | on Analysed | | | | |
| 1.13. | Screened | SP1 | Summary of Study Populations by Dose- Part A | By Dose and 'All Treatment' column<br>(Subjects on treatment except placebo)<br>should be included instead of 'Total'<br>column | SAC |
| 1.14. | Screened | SP1 | Summary of Study Populations by Cohort- Part A | By Cohort | SAC |
| 1.15. | Screened | SP1 | Summary of Study Populations by Dose- Part B | By Dose and 'All Treatment' column<br>(Subjects on treatment except placebo)<br>should be included instead of 'Total'<br>column | SAC |
| 1.16. | Screened | SP1 | Summary of Study Populations by Cohort- Part B | By Cohort | SAC |
| 1.17. | Screened | SP1 | Summary of Study Populations - Part C | By Dose and 'Total' column | SAC |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Demog | raphic and Bas | eline Characteris | tics | | , |
| 1.18. | Safety | DM3 | Summary of Demographic Characteristics - Part A | By cohort | SAC |
| 1.19. | Safety | DM1 | Summary of Demographic Characteristics - Part B | By cohort | SAC |
| 1.20. | Safety | DM3 | Summary of Demographic Characteristics - Part C | | SAC |
| 1.21. | Randomiz<br>ed | DM11 | Summary of Age Ranges – Part A | EudraCT, Disclosure display | SAC |
| 1.22. | Randomiz<br>ed | DM11 | Summary of Age Ranges – Part B | EudraCT, Disclosure display | SAC |
| 1.23. | Randomiz<br>ed | DM11 | Summary of Age Ranges – Part C | EudraCT, Disclosure display<br>Add 'Total' column | SAC |
| 1.24. | Safety | DM5 | Summary of Race and Racial Combinations - Part A | ICH E3, FDA, FDAAA, EudraCT,<br>Disclosure display<br>Add 'Total' column | SAC |
| 1.25. | Safety | DM5 | Summary of Race and Racial Combinations - Part B | ICH E3, FDA, FDAAA, EudraCT,<br>Disclosure display | SAC |
| 1.26. | Safety | DM5 | Summary of Race and Racial Combinations - Part C | ICH E3, FDA, FDAAA, EudraCT,<br>Disclosure display<br>Add 'Total' column | SAC |
| Prior an | d Concomitan | t Medications | | | |
| 1.27. | Safety | MH1 | Summary of Current/Past Medical Conditions - Part A | by Cohort | SAC |
| 1.28. | Safety | MH1 | Summary of Current/Past Medical Conditions - Part B | by Cohort | SAC |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.29. | Safety | MH1 | Summary of Current/Past Medical Conditions - Part C | By Cohort- since only one cohort,<br>'Total' column | SAC |
| 1.30. | Safety | CP_CM1 | Summary of Concomitant Medications - Part A | by Cohort | SAC |
| 1.31. | Safety | CP_CM1 | Summary of Concomitant Medications - Part B | by Cohort | SAC |
| 1.32. | Safety | CP_CM1 | Summary of Concomitant Medications - Part C | By Cohort- since only one cohort,<br>'Total' column | SAC |
| Exposur | e and Treatmen | t Compliance | | • | |
| 1.33. | Safety | EX1 | Summary of Exposure to Study Treatment - Part B | ICH E3 Dose and/or time on treatment, as applicable. Many possible considerations; defer to therapy area standards where available. For ClinPharm, a listing often substitutes for a table. | SAC |

# 13.12.5. Safety Tables

- The requirements for each display (i.e. IDSL, ICH, FDAAA etc) specified in the programming notes may be retained, all other red reference notes should be deleted.
- Select appropriate standard based on study design (i.e. parallel vs cross-over), when applicable.
- Suggested IDSL shells are noted in the third column, but other IDSL shells may be used, as appropriate

• The ADaM datasets for the Core Study Population/Safety displays can be found in the IDSL Library under Reference →Statistical Displays →ADaM Datasets for Core RAP Displays

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety | CP_AE1x | Summary of All Adverse Events by System Organ Class and Preferred Term - Part A | | SAC |
| 3.2. | Safety | CP_AE1p | Summary of All Adverse Events by System Organ Class and Preferred Term - Part B | | SAC |
| 3.3. | Safety | CP_AE1p | Summary of All Adverse Events by System Organ Class and Preferred Term by Study Phase - Part B | | SAC |
| 3.4. | Safety | CP_AE1x | Summary of All Adverse Events by System Organ Class and Preferred Term - Part C | | SAC |
| 3.5. | Safety | AE5B | Summary of All Adverse Events by Maximum Grade by System Organ Class and Preferred Term – Part A | | SAC |
| 3.6. | Safety | AE5B | Summary of All Adverse Events by Maximum Grade by System Organ Class and Preferred Term – Part B | | SAC |
| 3.7. | Safety | AE5B | Summary of All Adverse Events by Maximum Grade by System Organ Class and Preferred Term – Part C | | SAC |
| 3.8. | Safety | CP_AE1x | Summary All Drug-Related Adverse Events by System Organ<br>Class and Preferred Term- Part A | | SAC |
| 3.9. | Safety | CP_AE1p | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term - Part B | As 3.1 notes. | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10. | Safety | CP_AE1x | Summary All Drug-Related Adverse Events by System Organ<br>Class and Preferred Term - Part C | As 3.1 notes. | SAC |
| 3.11. | Safety | AE15 | Summary of Common (>=10%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) – Part A | FDAAA, EudraCT Disclosure display Common' to be defined by study/project team. For studies with very few events/participants, listing is sufficient: discuss this option with your disclosure representative. | SAC |
| 3.12. | Safety | AE15 | Summary of Common (>=10%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) – Part B | FDAAA, EudraCT Disclosure display 'Common' to be defined by study/project team. For studies with very few events/participants, listing is sufficient: discuss this option with your disclosure representative. | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.13. | Safety | AE15 | Summary of Common (>=10%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) – Part C | FDAAA, EudraCT Disclosure display 'Common' to be defined by study/project team. For studies with very few events/participants, listing is sufficient: discuss this option with your disclosure representative. | SAC |
| Serious | and Other Sig | nificant Advers | se Events | | |
| 3.14. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) - Part A | FDAAA, EudraCT By dose For studies with few events/participants listing is sufficient: discuss this option with your disclosure representative. | SAC |
| 3.15. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) - Part B | FDAAA, EudraCT For studies with few events/participants listing is sufficient: discuss this option with your disclosure representative. | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.16. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) - Part C | FDAAA, EudraCT For studies with few events/participants listing is sufficient: discuss this option with your disclosure representative. | SAC |
| Labora | tory: Chemistry | 1 | | | |
| 3.17. | Safety | LB1 | Summary of Clinical Chemistry Values – Part A | By dose Includes Baseline values. Includes pre-specified parameters repeated in conventional units. | SR, SAC |
| 3.18. | Safety | LB1 | Summary of Clinical Chemistry Values – Part B | By dose Includes Baseline values. Includes pre-specified parameters repeated in conventional units. | SR, SAC |
| 3.19. | Safety | LB1 | Summary of Clinical Chemistry Values – Part C | By treatment group (fed/fasted) Includes Baseline values. Includes pre-specified parameters repeated in conventional units. | SAC |
| 3.20. | Safety | LB1 | Summary of Chemistry Changes from Baseline - Part A | By dose and 'All Treatment' for all parameters mentioned in the protocol Includes Baseline values. Includes pre-specified parameters repeated in conventional units. | SR, SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.21. | Safety | LB1 | Summary of Chemistry Changes from Baseline - Part B | By dose for all parameters mentioned in the protocol Includes Baseline values. Includes pre-specified parameters repeated in conventional units. | SR, SAC |
| 3.22. | Safety | LB1 | Summary of Chemistry Changes from Baseline - Part C | By treatment group (fed/fasted) and 'Total' for all parameters mentioned in the protocol Includes Baseline values. Includes pre-specified parameters repeated in conventional units. | SAC |
| 3.23. | Safety | LB1 | Summary of Chemistry Percent Changes from Baseline - Part A | By dose and 'All Treatment' for all parameters mentioned in the protocol Includes Baseline values. Baseline values are required Includes pre-specified parameters repeated in conventional units. | SAC |
| 3.24. | Safety | LB1 | Summary of Chemistry Percent Changes from Baseline - Part B | By dose for all parameters mentioned in the protocol Includes Baseline values. Baseline values are required Includes pre-specified parameters repeated in conventional units. | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.25. | Safety | LB1 | Summary of Chemistry Percent Changes from Baseline - Part C | By treatment group (fed/fasted) and 'Total' for all parameters mentioned in the protocol Includes Baseline values. Baseline values are required Includes pre-specified parameters repeated in conventional units. | SAC |
| Labora | tory: Haematol | ogy | | | |
| 3.26. | Safety | LB1 | Summary of Haematology Values – Part A | By dose for all parameters mentioned in the protocol | SR, SAC |
| 3.27. | Safety | LB1 | Summary of Haematology Values – Part B | By dose for all parameters mentioned in the protocol | SR, SAC |
| 3.28. | Safety | LB1 | Summary of Haematology Values – Part C | By treatment group (fed/fasted) and<br>'Total' for all parameters mentioned in<br>the protocol | SAC |
| 3.29. | Safety | LB1 | Summary of Haematology Changes from Baseline - Part A | By dose and 'All Treatment' (treatment vs placebo) for all parameters mentioned in the protocol | SR, SAC |
| 3.30. | Safety | LB1 | Summary of Haematology Changes from Baseline - Part B | By dose for all parameters mentioned in the protocol | SR, SAC |
| 3.31. | Safety | LB1 | Summary of Haematology Changes from Baseline - Part C | By treatment group (fed/fasted) and<br>'Total' for all parameters mentioned in<br>the protocol | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.32. | Safety | LB1 | Summary of Haematology Percent Changes from Baseline - Part A | By dose and 'All Treatment' (treatment vs placebo) for all parameters mentioned in the protocol Baseline values are required | SAC |
| 3.33. | Safety | LB1 | Summary of Haematology Percent Changes from Baseline - Part B | By dose for all parameters mentioned in the protocol Baseline values are required | SAC |
| 3.34. | Safety | LB1 | Summary of Haematology Percent Changes from Baseline - Part C | By treatment group (fed/fasted) and 'Total' for all parameters mentioned in the protocol Baseline values are required | SAC |
| Hormo | ne Assessment | | | - | |
| 3.35. | Safety | LB1 | Summary of Hormone Assessment Values – Part B | By dose for all parameters mentioned in the protocol | SR, SAC |
| 3.36. | Safety | LB1 | Summary of Hormone Assessment Changes from Baseline - Part B | By dose for all parameters mentioned in the protocol | SR, SAC |
| 3.37. | Safety | LB1 | Summary of Hormone Assessment Percent Changes from Baseline - Part B | By dose for all parameters mentioned in the protocol Baseline values are required | SR, SAC |
| Labora | tory: Urinalysis | | | | |
| 3.38. | Safety | UR3b | Summary of Urinalysis Dipstick Results – Part A | ICH E3 Page by test Includes Baseline values. | SAC |
| 3.39. | Safety | UR3b | Summary of Urinalysis Dipstick Results – Part B | ICH E3 Page by test Includes Baseline values. | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.40. | Safety | UR3b | Summary of Urinalysis Dipstick Results – Part C | ICH E3 Page by testIncludes Baseline values. | SAC |
| Labora | tory: Liver Fund | ction | | | |
| 3.41. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting – Part A | IDSL | SAC |
| 3.42. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting – Part B | IDSL | SAC |
| 3.43. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting – Part C | IDSL | SAC |
| 3.44. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities – Part A | IDSL Listing may be sufficient if few events. | SAC |
| 3.45. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities – Part B | IDSL Listing may be sufficient if few events. | SAC |
| 3.46. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities – Part C | IDSL Listing may be sufficient if few events. | SAC |
| ECG | <b>'</b> | | | | 1 |
| 3.47. | Safety | EG1 | Summary of ECG Findings – Part A | IDSL As above for Chemistry, using ECG findings categories (and change from baseline categories, if applicable). | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.48. | Safety | EG1 | Summary of ECG Findings – Part B | IDSL As above for Chemistry, using ECG findings categories (and change from baseline categories, if applicable). | SAC |
| 3.49. | Safety | EG1 | Summary of ECG Findings – Part C | IDSL As above for Chemistry, using ECG findings categories (and change from baseline categories, if applicable). | SAC |
| 3.50. | Safety | EG2 | Summary of Change from Baseline in ECG Values – Part A | IDSL Includes Baseline values. | SAC |
| 3.51. | Safety | EG2 | Summary of Change from Baseline in ECG Values – Part B | IDSL<br>Includes Baseline values. | SAC |
| 3.52. | Safety | EG2 | Summary of Change from Baseline in ECG Values – Part C | IDSL<br>Includes Baseline values. | SAC |
| 3.53. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category – Part A | IDSL Recommended for studies with sufficiently large sample size or frequency of values of interest. | SAC |
| 3.54. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category – Part B | IDSL Recommended for studies with sufficiently large sample size or frequency of values of interest. | SAC |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.55. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category – Part C | IDSL Recommended for studies with sufficiently large sample size or frequency of values of interest. | SAC |
| 3.56. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category – Part A | IDSL Recommended for studies with sufficiently large sample size or frequency of values of interest. | SAC |
| 3.57. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category – Part B | IDSL Recommended for studies with sufficiently large sample size or frequency of values of interest. | SAC |
| 3.58. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category – Part C | IDSL Recommended for studies with sufficiently large sample size or frequency of values of interest. | SAC |
| Vital Si | gns | | | • | |
| 3.59. | Safety | VS1 | Summary of Vital Signs – Part A | ICH E3 Includes Baseline values. | SAC |
| 3.60. | Safety | VS1 | Summary of Vital Signs – Part B | ICH E3 Includes Baseline values. | SAC |
| 3.61. | Safety | VS1 | Summary of Vital Signs – Part C | ICH E3 Includes Baseline values. | SAC |
| 3.62. | Safety | VS1 | Summary of Change from Baseline in Vital Signs – Part A | ICH E3 Includes Baseline values. | SAC |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.63. | Safety | VS1 | Summary of Change from Baseline in Vital Signs – Part B | ICH E3 Includes Baseline values. | SAC |
| 3.64. | Safety | VS1 | Summary of Change from Baseline in Vital Signs – Part C | ICH E3<br>Includes Baseline values. | SAC |
| 3.65. | Safety | VS1 | Summary of Percent Change from Baseline in Vital Signs – Part A | ICH E3 Includes Baseline values. | SAC |
| 3.66. | Safety | VS1 | Summary of Percent Change from Baseline in Vital Signs – Part B | ICH E3 Includes Baseline values. | SAC |
| 3.67. | Safety | VS1 | Summary of Percent Change from Baseline in Vital Signs – Part C | ICH E3 Includes Baseline values. | SAC |

# 13.12.6. Safety Figures

- The requirements for each display (i.e. IDSL, ICH etc) specified in the programming notes may be retained, all other reference notes can be deleted.
- Select appropriate standard based on study design (i.e. parallel vs cross-over), when applicable.
- The ADaM datasets for the Core Study Population/Safety displays can be found in the IDSL Library under Reference → Statistical Displays → ADaM Datasets for Core RAP Displays.
| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Chemistry | / | | | |
| 3.1. | Safety | LB_PLOT1 | Individual Plot of Clinical Chemistry Parameters Over Time by Dose – Part A | By dose | SAC |
| 3.2. | Safety | LB_PLOT1 | Individual Plot of Clinical Chemistry Parameters Over Time by Dose – Part B | By dose | SAC |
| 3.3. | Safety | LB_PLOT1 | Individual Plot of Clinical Chemistry Parameters Over Time by Dose – Part C | By dose | SAC |
| 3.4. | Safety | LB_PLOT1 | Individual Plot of Clinical Chemistry Parameters Over Time by Subject – Part A | By subject | SAC |
| 3.5. | Safety | LB_PLOT1 | Individual Plot of Clinical Chemistry Parameters Over Time by Subject – Part C | By subject | SAC |
| 3.6. | Safety | LB_PLOT2 | Mean ±SD Plot of Change from Baseline for Clinical Chemistry Parameters Over Time by Dose – Part A | By dose and treatment (treatment vs placebo) for all parameters mentioned in the protocol | SAC |
| 3.7. | Safety | LB_PLOT2 | Mean ±SD Plot of Change from Baseline for Clinical Chemistry Parameters Over Time by Dose – Part B | By dose for all parameters mentioned in the protocol | SAC |
| 3.8. | Safety | LB_PLOT2 | Mean ±SD Plot of Change from Baseline for Clinical Chemistry Parameters Over Time by Dose – Part C | By treatment group (fed/fasted) for all parameters mentioned in the protocol | SAC |
| 3.9. | Safety | LB_PLOT2 | Mean ±SD Plot of Percent Change from Baseline for Clinical Chemistry Parameters Over Time by Dose – Part A | By dose and treatment (treatment vs placebo) for all parameters mentioned in the protocol | SAC |
| 3.10. | Safety | LB_PLOT2 | Mean ±SD Plot of Percent Change from Baseline for Clinical Chemistry Parameters Over Time by Dose – Part B | By dose for all parameters mentioned in the protocol | SAC |

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.11. | Safety | LB_PLOT2 | Mean ±SD Plot of Percent Change from Baseline for Clinical Chemistry Parameters Over Time by Dose – Part C | By treatment group (fed/fasted) for all parameters mentioned in the protocol | SAC |
| Labora | tory: Haematol | ogy | | | |
| 3.12. | Safety | LB_PLOT1 | Individual Plot of Haematology Parameters Over Time by Dose – Part A | By dose | SAC |
| 3.13. | Safety | LB_PLOT1 | Individual Plot of Haematology Parameters Over Time by Dose – Part B | By dose | SAC |
| 3.14. | Safety | LB_PLOT1 | Individual Plot of Haematology Parameters Over Time by Dose – Part C | | SAC |
| 3.15. | Safety | LB_PLOT1 | Individual Plot of Haematology Parameters Over Time by Subject – Part A | By Subject | SAC |
| 3.16. | Safety | LB_PLOT1 | Individual Plot of Haematology Parameters Over Time by Subject – Part C | By Subject | SAC |
| 3.17. | Safety | LB_PLOT2 | Mean ±SD Plot of Change from Baseline for Haematology<br>Parameters Over Time by Dose – Part A | By dose and treatment (treatment vs placebo) for all parameters mentioned in the protocol | SAC |
| 3.18. | Safety | LB_PLOT2 | Mean ±SD Plot of Change from Baseline for Haematology Parameters Over Time by Dose – Part B | By dose for all parameters mentioned in the protocol | SAC |
| 3.19. | Safety | LB_PLOT2 | Mean ±SD Plot of Change from Baseline for Haematology<br>Parameters Over Time by Dose – Part C | By treatment group (fed/fasted) for all parameters mentioned in the protocol | SAC |
| 3.20. | Safety | LB_PLOT2 | Mean ±SD Plot of Percent Change from Baseline for Haematology Parameters Over Time by Dose – Part A | By dose and treatment (treatment vs placebo) for all parameters mentioned in the protocol | SAC |

| Safety: | Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.21. | Safety | LB_PLOT2 | Mean ±SD Plot of Percent Change from Baseline for<br>Haematology Parameters Over Time by Dose – Part B | By dose for all parameters mentioned in the protocol | SAC |
| 3.22. | Safety | LB_PLOT2 | Mean ±SD Plot of Percent Change from Baseline for Haematology Parameters Over Time by Dose – Part C | By treatment group (fed/fasted) for all parameters mentioned in the protocol | SAC |
| Hormo | ne Assessment | | | , | |
| 3.23. | Safety | LB_PLOT1 | Individual Plot of Hormone Assessment Parameters Over Time by Dose – Part B | By dose | SAC |
| 3.24. | Safety | LB_PLOT2 | Mean ±SD Plot of Change from Baseline for Hormone<br>Assessment Parameters Over Time by Dose – Part B | By dose for all parameters mentioned in the protocol | SAC |
| 3.25. | Safety | LB_PLOT2 | Mean ±SD Plot of Percent Change from Baseline for Hormone<br>Assessment Parameters Over Time by Dose – Part B | By dose for all parameters mentioned in the protocol | SAC |
| Labora | tory: Liver Fun | ction | | | |
| 3.26. | Safety | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT – Part A | Recommended for larger studies, but not required for smaller studies. | SAC |
| 3.27. | Safety | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT – Part B | Recommended for larger studies, but not required for smaller studies. | SAC |

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.28. | Safety | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT – Part C | Recommended for larger studies, but not required for smaller studies. | SAC |

#### 13.12.7. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK con | centration | | | | |
| 4.1. | PK | PK01 | Summary of Plasma GSK3439171 Pharmacokinetic Concentration-Time Data (ng/mL) – Part A | | SAC |
| 4.2. | PK | PK01 | Summary of Plasma GSK3439171 Pharmacokinetic Concentration-Time Data (ng/mL) – Part B | | SAC |
| 4.3. | PK | PK01 | Summary of Plasma GSK3439171 Pharmacokinetic Concentration-Time Data (ng/mL) – Part C | | SAC |
| PK Urir | ne | | | | |
| 4.4. | PK | PK02 | Summary of Pharmacokinetic Urine Excretion Rate-Time Data – Part B | | SAC |
| PK deri | ved parameter | S | | | |
| 4.5. | PK | PK03 | Summary Statistics of Derived Plasma GSK3439171<br>Pharmacokinetic Parameters – Part A | | SAC |
| 4.6. | PK | PK03 | Summary Statistics of Derived Plasma GSK3439171<br>Pharmacokinetic Parameters – Part B | | SAC |
| 4.7. | PK | PK03 | Summary Statistics of Derived Plasma GSK3439171<br>Pharmacokinetic Parameters – Part C | | SAC |
| 4.8. | PK | PK05 | Summary Statistics of Log-Transformed Derived Plasma GSK3439171 Pharmacokinetic Parameters – Part A | | SAC |
| 4.9. | PK | PK05 | Summary Statistics of Log-Transformed Derived Plasma GSK3439171 Pharmacokinetic Parameters – Part B | | SAC |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.10. | PK | PK05 | Summary Statistics of Log-Transformed Derived Plasma<br>GSK3439171 Pharmacokinetic Parameters – Part C | | SAC |
| 4.11. | PK | PK_T1 | Statistical Analysis of Plasma GSK3439171 Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Part A | t1/2 | SAC |
| 4.12. | PK | PK_T1 | Statistical Analysis of Plasma GSK3439171 Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Part B | t1/2<br>Include 'Visit' as first column | SAC |
| 4.13. | PK | PK_T1 | Statistical Analysis of Plasma GSK3439171 Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Part C | t1/2 | SAC |
| 4.14. | PK | PK_T2 | Statistical Analysis of Log-Transformed Plasma GSK3439171 Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Part A | AUC(0-t), AUC(0-24), AUC(0-∞),<br>Cmax, Cτ, AUC(Rp) | SAC |
| 4.15. | PK | PK_T2 | Statistical Analysis of Log-Transformed Plasma GSK3439171 Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Part B | AUC(0- τ), AUC(0-∞), Cmax, Cτ Include 'Visit' as first column | SAC |
| 4.16. | PK | PK_T2 | Statistical Analysis of Log-Transformed Plasma GSK3439171 Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Part C | AUC(0-t), AUC(0-∞), Cmax | SAC |
| 4.17. | PK | PK_T5 | Statistical Analysis of Log-Transformed Plasma GSK3439171 Pharmacokinetic Parameters Assessing Accumulation Ratio and Time Invariance – Part B | | SAC |
| 4.18. | PK | PK_T6 | Statistical Analysis of Log-Transformed Plasma GSK3439171 Pharmacokinetic Parameters Assessing Achievement of Steady State – Part B | | SAC |

| Pharma | acokinetic: Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.19. | PK | PK_T3 | Statistical Analysis of Log-Transformed Plasma GSK3439171 Pharmacokinetic Parameters Assessing Dose Proportionality (Power Model) – Part A | AUC(0-t), AUC(0-∞) and Cmax | SAC |
| 4.20. | PK | PK_T4 | Statistical Analysis of Log-Transformed Plasma GSK3439171 Pharmacokinetic Parameters Assessing Dose Proportionality (Power Model) – Part B | AUC(0-τ) and Cmax By timepoint | SAC |
| Pharma | acogenetic | | | | |
| 4.21. | PK | GN1 | Summary of Subject Accountability – Part A | By cohort | SAC |
| 4.22. | PK | GN1 | Summary of Subject Accountability – Part B | | SAC |
| 4.23. | PK | GN1 | Summary of Subject Accountability – Part C | | SAC |
| 4.24. | PK | GN2 | Summary of Genetic Consent Not Obtained/Withdrawn – Part A | By cohort | SAC |
| 4.25. | PK | GN2 | Summary of Genetic Consent Not Obtained/Withdrawn – Part B | | SAC |
| 4.26. | PK | GN2 | Summary of Genetic Consent Not Obtained/Withdrawn – Part C | | SAC |

## 13.12.8. Pharmacokinetic Figures

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| ndivid | ual Concentrat | on Plots | | | <u> </u> |
| 4.1. | PK | PK16b | Individual Plasma GSK3439171 Concentration-time Plot (Linear and Semi-log) by Subject – Part A | | SAC |
| 4.2. | PK | PK16a | Individual Plasma GSK3439171 Concentration-time Plot (Linear and Semi-log) by Subject – Part B | | SAC |
| 4.3. | PK | PK16b | Individual Plasma GSK3439171 Concentration-time Plot (Linear and Semi-log) by Subject – Part C | | SAC |
| 4.4. | PK | PK24 | Individual Plasma GSK3439171 Concentration-time Plot (Linear and Semi-log) by Treatment – Part A | | SAC |
| 4.5. | PK | PK24 | Individual Plasma GSK3439171 Concentration-time Plot (Linear and Semi-log) by Treatment – Part B | | SAC |
| 4.6. | PK | PK24 | Individual Plasma GSK3439171 Concentration-time Plot (Linear and Semi-log) by Treatment – Part C | | SAC |
| 4.7. | PK | PK17 | Mean Plasma GSK3439171 Concentration-Time Plots (Linear and Semi-log) – Part A | | SAC |
| 4.8. | PK | PK17 | Mean Plasma GSK3439171 Concentration-Time Plots (Linear and Semi-log) – Part B | | SAC |
| 4.9. | PK | PK17 | Mean Plasma GSK3439171 Concentration-Time Plots (Linear and Semi-log) – Part C | | SAC |
| .10. | PK | PK18 | Median Plasma GSK3439171 Concentration-Time Plots (Linear and Semi-log) – Part A | | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.11. | PK | PK18 | Median Plasma GSK3439171 Concentration-Time Plots (Linear and Semi-log) – Part B | | SAC |
| 4.12. | PK | PK18 | Median Plasma GSK3439171 Concentration-Time Plots (Linear and Semi-log) – Part C | | SAC |
| 4.13. | PK | PK21 | Individual GSK3439171 Urine Excretion Rate-Time Plots (Linear and Semi-log) – Part B | | SAC |
| 4.14. | PK | PK22 | Mean GSK3439171 Urine Excretion Rate-Time Plots (Linear and Semi-log) – Part B | | SAC |
| 4.15. | PK | PK23 | Median GSK3439171 Urine Excretion Rate-Time Plots (Linear and Semi-log) – Part B | | SAC |

## 13.12.9. Pharmacodynamic (and / or Biomarker) Tables

| Pharma | Pharmacodynamic (and or Biomarker): Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Urinary | Urinary Tetranor and Urinary Creatinine | | | | |
| 6.1. | PD | PK03 | Summary Statistics of Urinary Tetranor and Urinary Creatinine<br>Concentration Data– Part A | | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.2. | PD | PK03 | Summary Statistics of Urinary Tetranor and Urinary Creatinine Parameters – Part A | PD parameters: tPGDM, tPGEM End points #: 1)Raw data (mass) 2)Creatinine corrected raw data, 3)Creatinine corrected aggregated data 0-12hrs, 4)Creatinine corrected aggregated data 12-24hrs 5)Creatinine corrected aggregated data 24-48hrs Baseline corrected value, Placebo corrected value and ratio of tPGDM/tPGEM for version 2,3 & 4 of the data mentioned above PD parameters: Creatinine End points #: 1)Raw data (mass), 2)Aggregated data 0-12hrs & 3)Aggregated data 12-24hrs 4) Aggregated data 24-48hrs Baseline corrected value and Placebo corrected value for version 2,3 & 4 of the data mentioned above | SAC |
| 6.3. | PD | PK03 | Summary Statistics of Urinary Tetranor and Urinary Creatinine<br>Concentration Data – Part B | | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.4. | PD | PK03 | Summary Statistics of Urinary Tetranor and Urinary Creatinine Parameters – Part B | PD parameters: tPGDM, tPGEM End points #: 1)Raw data (mass) 2)Creatinine corrected raw data, 3)Creatinine corrected aggregated data 0-12hrs, 4)Creatinine corrected aggregated data 12-24hrs 5)Creatinine corrected aggregated data 24-48hrs Baseline corrected value and ratio of tPGDM/tPGEM for version 3,4 & 5 of the data mentioned above PD parameters: Creatinine End points #: 1)Raw data (mass) 2)Aggregated data 0-12hrs & 3)Aggregated data 12-24hrs 4)Aggregated data 24-48hrs Baseline corrected value and Placebo corrected value for version 2,3 & 4 of the data mentioned above | SAC |

| Pharma<br>No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.5. | PD | PK05 | Summary Statistics of Log-Transformed Urinary Tetranor and Urinary Creatinine Parameters – Part A | PD parameters: tPGDM, tPGEM End points #: • 1)Raw data (mass) Predose aggregated data – 24-12hr, 12-0hr 2) Raw data (mass) Post dose aggregated data 0-12hrs, 12-24 hr & 24-48 hr 3)Creatinine corrected data predose aggregated – 24-12hr, 12-0hr 4)Creatinine corrected data postdose aggregated 0-12hrs, 12-24 hr & 24-48 PD parameters: Creatinine End points #: 1)Raw data (mass) Predose aggregated data – 24-12hr, 12-0hr 2) Raw data (mass) Post dose aggregated data 0-12hrs, 12-24 hr & 24-48 hr | SAC |

| Pharma | acodynamic (ar | nd or Biomarker): | Tables | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.6. | PD | PK05 | Summary Statistics of Log-Transformed Urinary Tetranor and Urinary Creatinine Parameters – Part B | PD parameters: tPGDM, tPGEM End points #: 1)Raw data (mass) Predose aggregated data – 24-12hr, 12-0hr 2) Raw data (mass) Post dose aggregated data 0-12hrs, 12-24 hr & 24-48 hr 3)Creatinine corrected data predose aggregated – 24-12hr, 12-0hr 4)Creatinine corrected data postdose aggregated 0-12hrs, 12-24 hr & 24-48 PD parameters: Creatinine End points #: 1)Raw data (mass) Predose aggregated data – 24-12hr, 12-0hr 2) Raw data (mass) Post dose aggregated data 0-12hrs, 12-24 hr & 24-48 hr | SAC |
| 6.7. | PD | PK05 | Summary Statistics of Muscle Concentration Data – Part B | | SAC |
| 6.8. | PD | PD_T1 | Statistical Analysis of Urinary Tetranor and Urinary Creatinine<br>Parameters: Mixed Effect Model – Part A | tPGDM, tPGEM, Creatinine,<br>Creatinine corrected tPGDM and<br>Creatinine corrected tPGEM | SAC |
| 6.9. | PD | PD_T1 | Statistical Analysis of Urinary Tetranor and Urinary Creatinine<br>Parameters: Mixed Effect Model – Part B | tPGDM, tPGEM, Creatinine,<br>Creatinine corrected tPGDM and<br>Creatinine corrected tPGEM | SAC |

# 13.12.10. Pharmacodynamic (and / or Biomarker) Figures

| Pharmaco | odynamic: Figi | ures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Urinary Te | tranor | | | | |
| 6.1. | PD | LB_PLOT1 | Plot of Urinary Tetranor and Urinary Creatinine vs Time by Dose– Part A | PD parameters: tPGDM, tPGEM End points #: • 1)Creatinine corrected raw data, 2)Creatinine corrected aggregated data 0-12hrs, 3)Creatinine corrected aggregated data 12-24hrs 4)Creatinine corrected aggregated data 24-48hrs • Baseline corrected value, Placebo corrected value and ratio of tPGDM/tPGEM for first 3 versions of the data mentioned above PD parameters: Creatinine End points #: • 1)Raw data, 2)Aggregated data 0-12hrs 3)Aggregated data 12-24hrs 4)Aggregated data 24-48hrs • Baseline corrected value and Placebo corrected value for first 3 versions of the data mentioned above Note: X-axis values – actual midpoint of collection | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.2. | PD | LB_PLOT1 | Plot of Urinary Tetranor and Urinary Creatinine vs Time by Dose– Part B | PD parameters: tPGDM, tPGEM for Day 1, 7, 9, 10 &17. End points #: 1)Creatinine corrected raw data, 2)Creatinine corrected aggregated data 0-12hrs, 3)Creatinine corrected aggregated data 12-24hrs 4)Creatinine corrected aggregated data 24-48hrs Baseline corrected value for first 3 versions of the data mentioned above PD parameters: Creatinine for Day 1, 7, 9, 10 &17 End points #: 1)Raw data, 2)Aggregated data 12-24hrs 4)Aggregated data 24-48hrs Baseline corrected value for first 3 versions of the data mentioned above Note1: X-axis values – actual midpoint of collection Note2: Panel plot each day as panel. Data available on day 1 for all cohorts, day 7 & 10 for cohort 3 only, day 9 &17 for cohort 1&2. | SAC |

| harmaco | odynamic: Figu | ıres | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 6.3. | PD | LB_PLOT1 | Plot of Urinary Tetranor and Urinary Creatinine vs Time by Subject– Part A | PD parameters: tPGDM, tPGEM End points #: 1)Creatinine corrected raw data, 2)Creatinine corrected aggregated data 0-12hrs, 3)Creatinine corrected aggregated data 12-24hrs 4)Creatinine corrected aggregated data 24-48hrs Baseline corrected value, Placebo corrected value and ratio of tPGDM/tPGEM for first 3 versions of the data mentioned above PD parameters: Creatinine End points #: 1)Raw data, 2)Aggregated data 0-12hrs & 3)Aggregated data 12-24hrs 4)Aggregated data 24-48hrs Baseline corrected value and Placebo corrected value for first 3 versions of the data mentioned above Note: X-axis values – actual midpoint of collection | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.4. | PD | LB_PLOT1 | Plot of Urinary Tetranor and Urinary Creatinine vs Time by Subject– Part B | PD parameters: tPGDM, tPGEM for Day 1, 7, 9, 10 &17 End points #: • 1)Creatinine corrected raw data, 2)Creatinine corrected aggregated data 0-12hrs, 3)Creatinine corrected aggregated data 12-24hrs 4)Creatinine corrected aggregated data 24-48hrs • Baseline corrected value for first 3 versions of the data mentioned above PD parameters: Creatinine for Day 1, 7, 9, 10 &17 End points #: • 1)Raw data, 2)Aggregated data 0-12hrs & 3)Aggregated data 12-24hrs 4)Aggregated data 24-48hrs • Baseline corrected value for first 3 versions of the data mentioned above Note1: X-axis values – actual midpoint of collection Note2: Each line(profile) for each day. Data available on day 1 for all cohorts, 7 & 10 for cohort 3 only, day 9 &17 for cohort 1&2. | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.5. | PD | LB_PLOT2 | Geometric mean and 95% CI Urinary Tetranor and Urinary Creatinine vs time – Part A | PD parameters: tPGDM, tPGEM End points #: • 1)Creatinine corrected raw data, 2)Creatinine corrected aggregated data 0-12hrs, 3)Creatinine corrected aggregated data 12-24hrs 4)Creatinine corrected aggregated data 24-48hrs • Baseline corrected value, Placebo corrected value and ratio of tPGDM/tPGEM for first 3 versions of the data mentioned above PD parameters: Creatinine End points #: • 1)Raw data, 2)Aggregated data 0-12hrs & 3)Aggregated data 12-24hrs 4)Aggregated data 24-48hrs • Baseline corrected value and Placebo corrected value for first 3 versions of the data mentioned above Note: X-axis values – planned midpoint of collection | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.6. | PD | LB_PLOT2 | Geometric mean and 95% CI Urinary Tetranor and Urinary Creatinine vs time – Part B | PD parameters: tPGDM, tPGEM for Day 1, 7, 9, 10 &17 End points #: • 1)Creatinine corrected raw data, 2)Creatinine corrected aggregated data 0-12hrs, 3)Creatinine corrected aggregated data 12-24hrs 4)Creatinine corrected aggregated data 24-48hrs • Baseline corrected value for first 3 versions of the data mentioned above PD parameters: Creatinine for Day 1, 7, 9, 10 &17 End points #: • 1)Raw data, 2)Aggregated data 0-12hrs & 3)Aggregated data 12-24hrs 4)Aggregated data 24-48hrs • Baseline corrected value for first 3 versions of the data mentioned above Note2: X-axis values – planned midpoint of collection Panel plot with each day as panel. Data available on day 1 for all cohorts, day 7 & 10 for cohort 3 only, day 9 &17 for cohort 1&2. | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| 6.7. | PD | LIVER14 | Plot of Urinary Tetranor and Urinary Creatinine vs PK Concentration by Dose– Part A | PD parameters: tPGDM and tPGEM End points #: | SAC |

| Pharmaco | Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.8. | PD | LIVER14 | Plot of Urinary Tetranor and Urinary Creatinine vs PK Concentration by Dose– Part B | PD parameters: tPGDM and Tpgem for Day 1, 10 &17 End points #: | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.9. | PD | LIVER14 | Plot of Urinary Tetranor and Urinary Creatinine vs PK<br>Concentration by Subject – Part A | PD parameters: tPGDM and tPGEM End points #: | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.10. | PD | LIVER14 | Plot of Urinary Tetranor and Urinary Creatinine vs PK Concentration by Subject – Part B | PD parameters: tPGDM and Tpgem for Day 1, 10 &17 End points #: | SAC |

| Pharmaco | odynamic: Fig | ures | | | |
|---|---|---|---|---|---|
| No. | Population IDSL / Example Shell Title Programming N | | Programming Notes | Deliverable<br>[Priority] | |
| 6.11. | PD | LB_PLOT1 | Plot of Ratio of Urinary Tetranor Parameters vs Time by Dose – Part A | Ratios of PD parameters to consider: tPGDM/tPGEM End points #: 1)Creatinine corrected data, 2)Creatinine corrected aggregated data 0-12hrs, 3)Creatinine corrected aggregated data 12-24hrs 4)Creatinine corrected aggregated data 24-48hrs Time matched ratio for above mentioned 4 versions of data Note: X-axis values – actual midpoint of collection | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.12. | PD | LB_PLOT1 | Plot of Ratio of Urinary Tetranor Parameters vs Time by Dose–<br>Part B | Ratios of PD parameters to consider: tPGDM/tPGEM for Day 1, 7, 9, 10 & 17 End points #: 1)Creatinine corrected raw data, 2)Creatinine corrected aggregated data 0-12hrs, 3)Creatinine corrected aggregated data 12-24hrs 4)Creatinine corrected aggregated data 24-48hrs Time matched ratio for above mentioned 4 versions of data Note: Panel plot with each panel for each day. Data available on day 1 for all cohorts, 7 & 10 for cohort 3 only, 9 &17 for cohort 1&2. | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| 6.13. | PD | LB_PLOT1 | Plot of Ratio of Urinary Tetranor Parameters vs Time by Subject– Part A | Ratios of PD parameters to consider: tPGDM/tPGEM End points #: 1)Creatinine corrected raw data, 2)Creatinine corrected aggregated data 0-12hrs, 3)Creatinine corrected aggregated data 12-24hrs 4)Creatinine corrected aggregated data 24-48hrs Time matched ratio for above mentioned 4 versions of data Note: X-axis values – actual midpoint of collection | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.14. | PD | LB_PLOT1 | Plot of Ratio of Urinary Tetranor Parameters vs Time by Subject– Part B | Ratios of PD parameters to consider: tPGDM/tPGEM for Day 1, 7, 9, 10 & 17 End points #: • 1)Creatinine corrected raw data, 2)Creatinine corrected aggregated data 0-12hrs, 3)Creatinine corrected aggregated data 12-24hrs 4)Creatinine corrected aggregated data 24-48hrs • Time matched ratio for above mentioned 4 versions of data Note: Each line(profile) for each day. Data available on day 1 for all cohorts, day 7 & 10 for cohort 3 only, day 9 &17 for cohort 1&2. | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| 6.15. | PD | LB_PLOT2 | Geometric mean and 95% CI Ratio of Urinary Tetranor Parameters vs time – Part A | Ratios of PD parameters to consider: tPGDM/tPGEM End points #: 1)Creatinine corrected raw data, 2)Creatinine corrected aggregated data 0-12hrs, 3)Creatinine corrected aggregated data 12-24hrs 4)Creatinine corrected aggregated data 24-48hrs Time matched ratio for above mentioned 4 versions of data Note: X-axis values – actual midpoint of collection | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.16. | PD | LB_PLOT2 | Geometric mean and 95% CI Ratio of Urinary Tetranor Parameters vs time – Part B | Ratios of PD parameters to consider: tPGDM/tPGEM for Day 1, 7, 9, 10 & 17 End points #: 1)Creatinine corrected raw data, 2)Creatinine corrected aggregated data 0-12hrs, 3)Creatinine corrected aggregated data 12-24hrs 4)Creatinine corrected aggregated data 24-48hrs Time matched ratio for above mentioned 4 versions of data Note: Panel plot with each panel for each day. Data available on day 1 for all cohorts, day 7 & 10 for cohort 3 only, day 9 &17 for cohort 1&2. | SAC |

#Refer to Section 10.1.1 for derivation of PD endpoints

#### 13.12.11. ICH Listings

- The requirements for each display (i.e. IDSL, ICH etc) specified in the programming notes may be retained, all other reference notes can be deleted.
- Select appropriate standard based on study design (i.e. parallel vs cross-over), when applicable.
- The ADaM datasets for the Core Study Population/Safety displays can be found in the IDSL Library under Reference → Statistical Displays → ADaM Datasets for Core RAP Displays.

| ICH: I | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subje | ect Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure – Part A | Journal Guidelines | SAC |
| 2. | Screened | ES7 | Listing of Reasons for Screen Failure – Part B | Journal Guidelines | SAC |
| 3. | Screened | ES7 | Listing of Reasons for Screen Failure – Part C | Journal Guidelines | SAC |
| 4. | Safety | CP_ES10x | Listing of Reasons for Study Withdrawal – Part A | ICH E3 | SAC |
| 5. | Safety | ES2 | Listing of Reasons for Study Withdrawal – Part B | ICH E3 | SAC |
| 6. | Safety | CP_ES10x | Listing of Reasons for Study Withdrawal – Part C | ICH E3 | SAC |
| 7. | Safety | SD2 | Listing of Reasons for Study Treatment Discontinuation – Part B | ICH E3 Required for all studies except single dose studies. | SAC |
| 8. | Safety | BL2 | Listing of Participants for Whom the Treatment Blind was Broken – Part A | ICH E3<br>Blinded studies only. | SAC |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 9. | Safety | BL1 | Listing of Participants for Whom the Treatment Blind was Broken – Part B | ICH E3 Blinded studies only. | SAC |
| 10. | Safety | BL2 | Listing of Participants for Whom the Treatment Blind was Broken – Part C | ICH E3 Blinded studies only. | SAC |
| 11. | Safety | TA2 | Listing of Planned and Actual Treatments – Part A | | SAC |
| 12. | Safety | TA1 | Listing of Planned and Actual Treatments – Part B | | SAC |
| 13. | Safety | TA2 | Listing of Planned and Actual Treatments – Part C | | SAC |
| Proto | col Deviations | | | | |
| 14. | Safety | DV2A | Listing of Important Protocol Deviations – Part A | ICH E3 Listing also includes analysis population exclusions. | SAC |
| 15. | Safety | DV2 | Listing of Important Protocol Deviations – Part B | ICH E3 Listing also includes analysis population exclusions. | SAC |
| 16. | Safety | DV2A | Listing of Important Protocol Deviations – Part C | ICH E3 Listing also includes analysis population exclusions. | SAC |
| 17. | Safety | IE4 | Listing of Participants with Inclusion/Exclusion Criteria Deviations – Part A | ICH E3 | SAC |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 18. | Safety | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations – Part B | ICH E3 | SAC |
| 19. | Safety | IE4 | Listing of Participants with Inclusion/Exclusion Criteria Deviations – Part C | ICH E3 | SAC |
| Popu | lations Analys | ed | | | |
| 20. | Randomized | SP3a | Listing of Participants Excluded from Any Population – Part A | e.g., participants screened but not randomized, participants randomized but not treated, participants with deviations leading to exclusion from per protocol population (can be separate listing per population). | SAC |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 21. | Randomized | SP3 | Listing of Participants Excluded from Any Population – Part B | ICH E3 e.g., participants screened but not randomized, participants randomized but not treated, participants with deviations leading to exclusion from per protocol population (can be separate listing per population). | SAC |
| 22. | Randomized | SP3a | Listing of Participants Excluded from Any Population – Part C | ICH E3 e.g., participants screened but not randomized, participants randomized but not treated, participants with deviations leading to exclusion from per protocol population (can be separate listing per population). | SAC |
| Dem | ographic and B | aseline Chara | cteristics | <b>'</b> | 1 |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 23. | Safety | DM4 | Listing of Demographic Characteristics – Part A | ICH E3 | SAC |
| 24. | Safety | DM2 | Listing of Demographic Characteristics – Part B | ICH E3 | SAC |
| 25. | Safety | DM4 | Listing of Demographic Characteristics – Part C | ICH E3 | SAC |
| 26. | Safety | SU2 | Listing of Substance Use – Part A | | SAC |
| 27. | Safety | SU2 | Listing of Substance Use – Part B | | SAC |
| 28. | Safety | SU2 | Listing of Substance Use – Part C | | SAC |
| Prior | and Concomit | ant Medicatio | ns | | |
| 29. | Safety | CP_CM4 | Listing of Concomitant Medications Using Generic Term – Part A | | SAC |
| 30. | Safety | CP_CM3 | Listing of Concomitant Medications Using Generic Term – Part B | | SAC |
| 31. | Safety | CP_CM4 | Listing of Concomitant Medications Using Generic Term – Part C | | SAC |
| 32. | Safety | MH3 | Listing of Medical Conditions – Part A | | SAC |
| 33. | Safety | MH2 | Listing of Medical Conditions – Part B | | SAC |
| 34. | Safety | MH3 | Listing of Medical Conditions – Part C | | SAC |
| 35. | Safety | FH5 | Listing of Family History Conditions – Part A | | SAC |
| 36. | Safety | FH5 | Listing of Family History Conditions – Part B | | SAC |
| 37. | Safety | FH5 | Listing of Family History Conditions – Part C | | SAC |
| Expo | sure and Treat | ment Complia | ince | | |
| 38. | Safety | EX4 | Listing of Exposure Data – Part A | ICH E3 | SAC |
| 39. | Safety | EX3 | Listing of Exposure Data – Part B | ICH E3 | SAC |
| 40. | Safety | EX4 | Listing of Exposure Data – Part C | ICH E3 | SAC |
| Adve | erse Events | | | | |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 41. | Safety | CP_AE9 | Listing of All Adverse Events – Part A | ICH E3 | SAC |
| 42. | Safety | CP_AE8 | Listing of All Adverse Events – Part B | ICH E3 | SAC |
| 43. | Safety | CP_AE9 | Listing of All Adverse Events – Part C | ICH E3 | SAC |
| 44. | Safety | CP_AE9 | Listing of Drug Related Adverse Events – Part A | ICH E3 Fatal and Non-Fatal SAEs are combined into a single listing for ClinPharm studies (i.e., "Listing of Serious Adverse Events"). | SAC |
| 45. | Safety | CP_AE8 | Listing of Drug Related Adverse Events – Part B | ICH E3 Fatal and Non-Fatal SAEs are combined into a single listing for ClinPharm studies (i.e., "Listing of Serious Adverse Events"). | SAC |
| ICH: | CH: Listings | | | | | | | | | |
|---|---|---|---|---|---|--|--|--|--|--|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | | | | | |
| 46. | Safety | CP_AE9 | Listing of Drug Related Adverse Events – Part C | ICH E3 Fatal and Non-Fatal SAEs are combined into a single listing for ClinPharm studies (i.e., "Listing of Serious Adverse Events"). | SAC | | | | | |
| 47. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events – Part A | ICH E3 | SAC | | | | | |
| 48. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events – Part B | ICH E3 | SAC | | | | | |
| 49. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events – Part C | ICH E3 | SAC | | | | | |
| 50. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text – Part A | IDSL | SAC | | | | | |
| 51. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text – Part B | IDSL | SAC | | | | | |
| 52. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text – Part C | IDSL | SAC | | | | | |
| Serio | us and Other S | Significant Adv | verse Events | | | | | | | |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 53. | Safety | CP_AE9a | Listing of Serious Adverse Events (Fatal & Non-Fatal) – Part A | ICH E3 Fatal and Non-Fatal SAEs are combined into a single listing for ClinPharm studies (i.e., "Listing of Serious Adverse Events"). | SAC |
| 54. | Safety | CP_AE8a | Listing of Serious Adverse Events (Fatal & Non-Fatal) – Part B | ICH E3 Fatal and Non-Fatal SAEs are combined into a single listing for ClinPharm studies (i.e., "Listing of Serious Adverse Events"). | SAC |
| 55. | Safety | CP_AE9a | Listing of Serious Adverse Events (Fatal & Non-Fatal) – Part C | ICH E3 Fatal and Non-Fatal SAEs are combined into a single listing for ClinPharm studies (i.e., "Listing of Serious Adverse Events"). | SAC |
| 56. | Safety | CP_AE9 | Listing of Adverse Events Leading to Withdrawal from Study – Part A | ICH E3 | SAC |
| 57. | Safety | CP_AE8 | Listing of Adverse Events Leading to Withdrawal from Study – Part B | ICH E3 | SAC |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 58. | Safety | CP_AE9 | Listing of Adverse Events Leading to Withdrawal from Study – Part C | ICH E3 | SAC |
| Liver | events | | | | |
| 59. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting – Part A | IDSL | SAC |
| 60. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting – Part B | IDSL | SAC |
| 61. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting – Part C | IDSL | SAC |
| 62. | Safety | LIVER7 | Listing of Liver Biopsy Details – Part A | | SAC |
| 63. | Safety | LIVER7 | Listing of Liver Biopsy Details – Part B | | SAC |
| 64. | Safety | LIVER7 | Listing of Liver Biopsy Details – Part C | | SAC |
| 65. | Safety | LIVER8 | Listing of Liver Imaging Details – Part A | | SAC |
| 66. | Safety | LIVER8 | Listing of Liver Imaging Details – Part B | | SAC |
| 67. | Safety | LIVER8 | Listing of Liver Imaging Details – Part C | | SAC |
| All La | aboratory | | | | |
| 68. | Safety | LB14 | Listing of Clinical Chemistry Laboratory Data with Character Results – Part A | ICH E3 | SAC |
| 69. | Safety | LB14 | Listing of Clinical Chemistry Laboratory Data with Character Results – Part B | ICH E3 | SAC |
| 70. | Safety | LB14 | Listing of Clinical Chemistry Laboratory Data with Character Results – Part C | ICH E3 | SAC |
| 71. | Safety | CP_LB6 | Listing of All Clinical Chemistry Laboratory Data for Subjects with PCI Abnormalities – Part A | Add 'Lab test' column<br>before 'Treatment/Period'<br>column' | SAC |
| 72. | Safety | CP_LB5 | Listing of All Clinical Chemistry Laboratory Data for Subjects with PCI Abnormalities – Part B | Add 'Lab test' column<br>before 'Treatment/Period'<br>column' | SAC |

| ICH: | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 73. | Safety | CP_LB6 | Listing of All Clinical Chemistry Laboratory Data for Subjects with PCI Abnormalities – Part C | Add 'Lab test' column<br>before 'Treatment/Period'<br>column' | SAC |
| 74. | Safety | CP_LB6 | Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance – Part A | Add 'Lab test' column<br>before 'Treatment/Period'<br>column' | SAC |
| 75. | Safety | CP_LB5 | Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance – Part B | Add 'Lab test' column<br>before 'Treatment/Period'<br>column' | SAC |
| 76. | Safety | CP_LB6 | Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance – Part C | Add 'Lab test' column<br>before 'Treatment/Period'<br>column' | SAC |
| 77. | Safety | LB14 | Listing of Haematology Laboratory Data with Character Results – Part A | ICH E3 'Treatment/Period' will be included as column and will be added after 'Lab Test' | SAC |
| 78. | Safety | LB14 | Listing of Haematology Laboratory Data with Character Results – Part B | ICH E3 | SAC |
| 79. | Safety | LB14 | Listing of Haematology Laboratory Data with Character Results – Part C | ICH E3 | SAC |
| 80. | Safety | CP_LB6 | Listing of All Haematology Laboratory Data for Subjects with PCI Abnormalities – Part A | Add 'Lab test' column<br>before 'Treatment/Period'<br>column' | SAC |
| 81. | Safety | CP_LB5 | Listing of All Haematology Laboratory Data for Subjects with PCI Abnormalities – Part B | Add 'Lab test' column<br>before 'Treatment/Period'<br>column' | SAC |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 82. | Safety | CP_LB6 | Listing of All Haematology Laboratory Data for Subjects with PCI Abnormalities – Part C | Add 'Lab test' column<br>before 'Treatment/Period'<br>column' | SAC |
| 83. | Safety CP_LB6 Listing of Haematology Abnormalities of Potential Clinical Importance – Part A be | | Add 'Lab test' column<br>before 'Treatment/Period'<br>column' | SAC | |
| 84. | Safety | CP_LB5 | Listing of Haematology Abnormalities of Potential Clinical Importance – Part B | Add 'Lab test' column<br>before 'Treatment/Period'<br>column' | SAC |
| 85. | Safety | CP_LB6 | Listing of Haematology Abnormalities of Potential Clinical Importance – Part C | Add 'Lab test' column<br>before 'Treatment/Period'<br>column' | SAC |
| 86. | Safety | LB14 | Listing of Hormone Assessment Data with Character Results – Part B | ICH E3 | SAC |
| 87. | Safety | LB14 | Listing of Urinalysis Data with Character Results – Part A | ICH E3 | SAC |
| 88. | Safety | LB14 | Listing of Urinalysis Laboratory Data with Character Results – Part B | ICH E3 | SAC |
| 89. | Safety | LB14 | Listing of Urinalysis Laboratory Data with Character Results – Part C | ICH E3 | SAC |
| 90. | Safety | UR2B | Listing of Urinalysis Data for Participants with Any Value of Potential Clinical Importance – Part A | ICH E3 Display ALL data for a subject who experienced a value of potential clinical importance. | SAC |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 91. | Safety | UR2A | Listing of Urinalysis Data for Participants with Any Value of Potential Clinical Importance – Part B | ICH E3 Display ALL data for a subject who experienced a value of potential clinical importance. | SAC |
| 92. | Safety | UR2B | Listing of Urinalysis Data for Participants with Any Value of Potential Clinical Importance – Part C | ICH E3 Display ALL data for a subject who experienced a value of potential clinical importance. | SAC |
| ECG | | | | 1 | |
| 93. | Safety | CP_EG4 | Listing of All ECG Values for Subjects with any Value of Potential Clinical Importance – Part A | IDSL Required for ClinPharm studies only. Display ALL ECGs for a subject who experienced a value of potential clinical importance. | SAC |

| ICH: | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 94. | Safety | CP_EG3 | Listing of All ECG Values for Subjects with any Value of Potential Clinical Importance – Part B | IDSL Required for ClinPharm studies only. Display ALL ECGs for a subject who experienced a value of potential clinical importance. | SAC |
| 95. | Safety | CP_EG4 | Listing of All ECG Values for Subjects with any Value of Potential Clinical Importance – Part C | IDSL Required for ClinPharm studies only. Display ALL ECGs for a subject who experienced a value of potential clinical importance. | SAC |
| 96. | Safety | CP_EG4 | Listing of ECG Values of Potential Clinical Importance – Part A | IDSL<br>Required for<br>ClinPharm studies<br>only. | SAC |
| 97. | Safety | CP_EG3 | Listing of ECG Values of Potential Clinical Importance – Part B | IDSL Required for ClinPharm studies only. | SAC |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 98. | Safety | CP_EG4 | Listing of ECG Values of Potential Clinical Importance – Part C | IDSL<br>Required for<br>ClinPharm studies<br>only. | SAC |
| 99. | Safety | CP_EG6 | Listing of All ECG Findings for Subjects with an Abnormal Finding – Part A | | SAC |
| 100. | Safety | CP_EG5 | Listing of All ECG Findings for Subjects with an Abnormal Finding – Part B | | SAC |
| 101. | Safety | CP_EG6 | Listing of All ECG Findings for Subjects with an Abnormal Finding – Part C | | SAC |
| 102. | Safety | CP_EG6 | Listing of Abnormal ECG Findings – Part A | IDSL Required for ClinPharm studies only. | SAC |
| 103. | Safety | CP_EG5 | Listing of Abnormal ECG Findings – Part B | IDSL Required for ClinPharm studies only. | SAC |
| 104. | Safety | CP_EG6 | Listing of Abnormal ECG Findings – Part C | IDSL Required for ClinPharm studies only. | SAC |
| Vital | Signs | | | | |

| ICH: | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 105. | Safety | CP_VS5 | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance – Part A | IDSL Required for ClinPharm studies only. Display ALL Vital Signs for a subject who experienced a value of potential clinical importance. | SAC |
| 106. | Safety | CP_VS4 | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance – Part B | IDSL Required for ClinPharm studies only. Display ALL Vital Signs for a subject who experienced a value of potential clinical importance. | SAC |
| 107. | Safety | CP_VS5 | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance – Part C | IDSL Required for ClinPharm studies only. Display ALL Vital Signs for a subject who experienced a value of potential clinical importance. | SAC |

| ICH: I | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 108. | Safety | CP_VS5 | Listing of Vital Signs of Potential Clinical Importance – Part A | IDSL<br>Required for<br>ClinPharm studies<br>only. | SAC |
| 109. | Safety | CP_VS4 | Listing of Vital Signs of Potential Clinical Importance – Part B | IDSL Required for ClinPharm studies only. | SAC |
| 110. | Safety | CP_VS5 | Listing of Vital Signs of Potential Clinical Importance – Part C | IDSL Required for ClinPharm studies only. | SAC |

# 13.12.12. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acokinetics | | | | |
| 111. | PK | PK08 | Listing of Plasma GSK3439171 Pharmacokinetic Concentration (ng/mL) - Time Data – Part A | | SAC |
| 112. | PK | PK07 | Listing of Plasma GSK3439171 Pharmacokinetic Concentration (ng/mL) - Time Data – Part B | | SAC |
| 113. | PK | PK08 | Listing of Plasma GSK3439171 Pharmacokinetic Concentration (ng/mL) - Time Data – Part C | | SAC |
| 114. | PK | PK09 | Listing of Urine Sample Collections – Part B | | SAC |
| 115. | PK | PK11 | Listing of Urine Excretion Rate Data – Part B | | SAC |
| 116. | PK | PK14 | Listing of Derived Plasma GSK3439171 Pharmacokinetic Parameters – Part A | | SAC |
| 117. | PK | PK13 | Listing of Derived Plasma GSK3439171 Pharmacokinetic Parameters – Part B | | SAC |
| 118. | PK | PK14 | Listing of Derived Plasma GSK3439171 Pharmacokinetic Parameters – Part C | | SAC |
| 119. | PK | NA | Raw SAS Output from Statistical Analysis plasma GSK3439171 Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Part A | | SAC |
| 120. | PK | NA | Raw SAS Output from Statistical Analysis plasma GSK3439171 Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Part B | | SAC |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 121. | PK | NA | Raw SAS Output from Statistical Analysis plasma GSK3439171<br>Pharmacokinetic Parameters: Analysis of Variance (ANOVA) –<br>Part C | | SAC |
| 122. | PK | NA | Raw SAS Output from Statistical Analysis of Log Transformed plasma GSK3439171 Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Part A | | SAC |
| 123. | PK | NA | Raw SAS Output from Statistical Analysis of Log Transformed plasma GSK3439171 Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Part B | | SAC |
| 124. | PK | NA | Raw SAS Output from Statistical Analysis of Log Transformed plasma GSK3439171 Pharmacokinetic Parameters: Analysis of Variance (ANOVA) – Part C | | SAC |
| 125. | PK | NA | Raw SAS Output from Statistical Analysis of Log-Transformed Plasma GSK3439171 Pharmacokinetic Parameters Assessing Accumulation Ratio – Part B | | SAC |
| | PK | NA | Raw SAS Output from Statistical Analysis of Log-Transformed Plasma GSK3439171 Pharmacokinetic Parameters Assessing Time Invariance – Part B | | SAC |
| 126. | PK | NA | Raw SAS Output from Statistical Analysis of Log-Transformed Plasma GSK3439171 Pharmacokinetic Parameters Assessing Achievement of Steady State – Part B | | SAC |
| 127. | PK | NA | Raw SAS Output from Statistical Analysis of log transformed plasma GSK3439171 Pharmacokinetic Parameters Assessing Dose Proportionality (Power Model) – Part A | | SAC |

| Non-ICI | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 128. | PK | NA | Raw SAS Output from Statistical Analysis of log transformed plasma GSK3439171 Pharmacokinetic Parameters Assessing Dose Proportionality (Power Model) – Part B | | SAC |
| 129. | PK | | Listing of Entero-Test – Part B | | SAC |
| Pharma | codynamics/B | iomarkers | | | |
| 130. | PD | PD_L1 | Listing of All Pharmacodynamic Parameters – Part A | | SAC |
| 131. | PD | PD_L1 | Listing of Urine Pharmacodynamic Parameters – Part B | | SAC |
| 132. | PD | PD_L1 | Listing of Muscle Pharmacodynamic Parameters – Part B | | SAC |
| 133. | PD | NA | Raw SAS Output from Statistical Analysis of Log Transformed Pharmacodynamic Parameters: Analysis of Variance (ANOVA) – Part A | | SAC |
| 134. | PD | NA | Raw SAS Output from Statistical Analysis of Log Transformed Pharmacodynamic Parameters: Analysis of Variance (ANOVA) – Part B | | SAC |

# 13.12.13. Other Listings

| Other Listings | | | | | |
|---|---|---|---|---|---|
| No. Population IDSL / Example Shell | | | Title | Programming Notes | Deliverable<br>[Priority] |
| Study Population Tables | | | | | |
| 135. | Screened | OT_L1 | Listing of Rescreened Subjects | | SAC |

## 13.13. Example Mock Shells for Data Displays

Please note that the mock shells provided below are not study specific but example mock shells.

Example LB\_PLOT1

Protocol: XYZ100001 Page 1 of 1

Population: Safety/Other study specific

Figure 8.xx

### Individual Plot of Clinical Chemistry Parameters Over Time by Dose – Part A



Please add lower and upper normal ranges in the plot.

Page 1 of 1

Example LB\_PLOT2
Protocol: XYZ100001

Population: Safety/Other study specific

Figure 8.xx

Mean  $\pm \text{SD}$  Plot of Change from Baseline for Clinical Chemistry Parameters Over time - Part A




Example : PK\_T1
Protocol : GSKxxx

Population : Pharmacokinetic

Table PK\_T1
Statistical Analysis of plasma GSKxxx Pharmacokinetic Parameters: ANOVA – Part A

| Parameter | Treatment | N | n | LS Mean | 95% CI<br>(Lower,Upper) | {%CVw} |
|---|---|---|---|---|---|---|
| AUC(0-t) (units) | ) 50mg | 24 | 24 | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xx |
| | 100mg | 24 | 24 | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XX |
| | 200mg | 24 | 24 | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XX |
| Cmax (units) | 50mg | 24 | 24 | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XX |
| | 100mg | 24 | 24 | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XX |
| | 200mg | 24 | 24 | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XX |


Example : PK\_T2 Protocol : GSKxxx

Population: Pharmacokinetic

Table PK\_T2
Statistical Analysis of log transformed plasma GSKxxx Pharmacokinetic Parameters: ANOVA – Part A

| Parameter | Treatment | N | n | LS Geom.<br>Mean | 95% CI<br>(Lower,Upper) | {%CVw} |
|---|---|---|---|---|---|---|
| AUC(0-t) (units) | 50mg | 24 | 24 | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xx |
| | 100mg | 24 | 24 | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XX |
| | 200mg | 24 | 24 | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XX |
| Cmax (units) | 50mg | 24 | 24 | XXXX.XX | (xxxx.xx,xxxx.xx) | xx.xx |
| | 100mg | 24 | 24 | XXXX.XX | (xxxx.xx,xxxx.xx) | xx.xx |
| | 200mg | 24 | 24 | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XX |

Example: PK\_T3

Protocol : GSKxxx

Population: Pharmacokinetic

Table PK\_T3
Statistical Analysis of log transformed plasma GSKxxx Pharmacokinetic Parameters Assessing Dose Proportionality
(Power Model) - Part A

| Parameter (units) | Slope | 90% CI of the Slope |
|---------------------------|---------------------------|---------------------|
| | Log Parameter vs Log Dose | |
| AUC(0-t) (μg.h/mL) | X.XX | (x.xxx, x.xxx) |
| $AUC(0-\infty)$ (µg.h/mL) | X.XX | (x.xxx, x.xxx) |
| $AUC(0-\tau)$ (µg.h/mL) | X.XX | (x.xxx, x.xxx) |


Example : PK\_T4
Protocol : GSKxxx

Population : Pharmacokinetic

Table PK\_T4
Statistical Analysis of log transformed plasma GSKxxx Pharmacokinetic Parameters Assessing Dose Proportionality
(Power Model) – Part B

| Visit | Parameter (units) | Slope | 90% CI of the Slope |
|---|---|---|---|
| | | Log Parameter vs Log Dose | |
| Day 1 | AUC(0-t) (μg.h/mL) | X.XX | (x.xxx, x.xxx) |
| | $AUC(0-\infty)$ (µg.h/mL) | X.XX | (x.xxx, x.xxx) |
| | $AUC(0-\tau)$ (µg,h/mL) | X.XX | (x.xxx, x.xxx) |

Example : PK\_T5
Protocol : GSKxxx Page 1 of n

Population: Pharmacokinetic

### Table PK\_T5

Statistical Analysis of log transformed plasma GSKxxx Pharmacokinetic Parameters Assessing Accumulation Ratio and Time Invariance – Part B

| Freatment | Parameter (units) | Compa | rison | 1 Geom.LsMean | | Ratio | | 90%<br>Confidence Interval | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | n | Test | n Ref | | Confidence | e miervar |
| XXmg | AUC(Ro)(µg.h/mL) | Day 17 vs Da | y 1 | XX | x.xxx | xx x.xxx | x.xxx | ( x.xxx, | x.xxx ) |
| | Cmax(RCmax)(µg/mL) | Day 17 vs Da | y 1 | XX | x.xxx | xx x.xxx | x.xx | ( x.xxx, | ж.жжж ) |
| | AUC (Res ) (ug.h/mL) | Dav 17 vs Da | v 1 | XX | x.xxx | XX X.XXX | x.xxx | ( x.xxx. | x.xxx ) |

Example: PK\_T6

Protocol : GSKxxx

Population: Pharmacokinetic

Table PK\_T6

Statistical Analysis of log transformed plasma GSKxxx Pharmacokinetic Parameters Assessing Achievement of Steady State–Part B

| Parameter | Treatment | Day | Back-Transformed Slope | 90% Confidence Interval |
|---|---|---|---|---|
| Ctrough | xxmg | 1-17 | K. KKK | (x.xxx, x.xxx) |
| | xxmg | 1-17 | x.xxx | (x.xxx, x.xxx) |

•

•

.

Example: PD\_T1 Page 1 of n

Example : PD\_T1
Protocol : GSKxxx

Population : Pharmacodynamic

Table

Statistical Analysis of Urinary Tetranor and Urinary Creatinine Parameters:

Mixed Effect Model - Part A

| Parameter: tPGE | EM | | | |
|---|---|---|---|---|
| Visit | | Placebo<br>(N=xxx) | Dose1(N=xxx) | Dose6<br>(N=xxx) |
| Day -1, 24-12hr | n Adjusted Geometric Mean 90% C.I. | xxx<br>x.xxx<br>(x.xxx, x.xxx) | xxx<br>x.xxx<br>(x.xxx, x.xxx) | xxx<br>x.xxx<br>(x.xxx, x.xxx) |
| Day -1, 12-0hr | n<br>Adjusted Geometric Mean<br>90% C.I. | xxx<br>x.xxx<br>(x.xxx, x.xxx) | xxx<br>x.xxx<br>(x.xxx, x.xxx) | xxx<br>x.xxx<br>(x.xxx, x.xxx) |
| Day 1, 0-12hr | n<br>Adjusted Geometric Mean<br>90% C.I. | xxx<br>x.xxx<br>(x.xxx, x.xxx) | xxx<br>x.xxx<br>(x.xxx, x.xxx) | xxx<br>x.xxx<br>(x.xxx, x.xxx) |
| | Change from Baseline 90% C.I. | x.xxx<br>(x.xxx, x.xxx) | x.xxx<br>(x.xxx, x.xxx) | x.xxx<br>(x.xxx, x.xxx) |
| Day 1, 12-24hr | n<br>Adjusted Geometric Mean<br>90% C.I. | xxx<br>x.xxx<br>(x.xxx, x.xxx) | xxx<br>x.xxx<br>(x.xxx, x.xxx) | xxx<br>x.xxx<br>(x.xxx, x.xxx) |

#### CONFIDENTIAL

209275

| | Change from Baseline | X.XXX | X.XXX | X.XXX |
|---|---|---|---|---|
| | 90% C.I. | (x.xxx, x.xxx) | (x.xxx, x.xxx) | (x.xxx, x.xxx) |
| Day 1, 24-48hr | n | XXX | XXX | XXX |
| | Adjusted Geometric Mean | x.xxx | x.xxx | x.xxx |
| | 90% C.I. | (x.xxx, x.xxx) | (x.xxx, x.xxx) | (x.xxx, x.xxx) |

Example OT\_L1

Protocol : GSKxxx Population : Screened

Listing 11 Listing of Re-screened Subjects

| Part | Unique Subject<br>Id. | First Screening<br>Number | Second<br>Screening<br>Number |
|---|---|---|---|
| Part A | xxxxxx.xxxxxx | xxxxx | xxxxx |
| | XXXXXX.XXXXXX | XXXXXX | XXXXXX |
| | XXXXXX.XXXXXX | XXXXXX | XXXXXX |